

### Studienprotokoll

# Kohortenstudie zu pflanzenbasierter Ernährung <a href="CO">CO</a>hort on <a href="PLANT">PLANT</a>-based Diets (COPLANT) Study



#### Inhalt

| 1. | . Н | tergrund | |
|---|---|---|---|
| 2. | . W | issenschaftliche Ziele der COPLANT-Studie | |
| 3. | . S | Studienzentren, assoziierte Partner und Verantwortlichkeiten | |
| 4. | . Projektkoordination | | |
| 5. | . S | tudiendesign | 12 |
| | 5.1 | Studientyp | 12 |
| | 5.2 | Ein- und Ausschlusskriterien | 13 |
| | 5.3 | Rekrutierung der Studienteilnehmenden | 14 |
| | 5.4 | Zeitplan | 15 |
| 6. | . В | asiserhebung | 16 |
| | 6.1 | Ablauf der Basiserhebung | 16 |
| | 6.2 | Erhebung der Ernährungsweise | 18 |
| | 6.3 | Anthropometrie | 22 |
| | 6.4 | Bioelektrische Impedanzanalyse | 22 |
| | 6.5 | Messung der Knochengesundheit | 22 |
| | 6.6 | Blutdruckmessung | 22 |
| | 6.7 | Akzelerometrie | 23 |
| | 6.8 | Messung der Handgreifkraft | 23 |
| | 6.9 | Weitere Untersuchungen | 23 |
| | 6.10 | Erhebung der Einnahme von Arzneimitteln und Nahrungsergänzungsmitteln | 23 |
| | 6.11 | Befragungen | 23 |
| | 6.12 | Sammlung von biologischen Proben | 24 |
| 7. | . N | achbeobachtung | 25 |
| 8. | . S | tatistische Datenanalyse | 26 |
| | 8.1 | Statistische Methoden | 26 |
| | 8.2 | Planung des Stichprobenumfanges | 27 |
| 9. | . N | achhaltigkeitsanalyse | 29 |
| 1( | 0. M | odul "Schwangere und Stillende" | 30 |

| 10.1 | Wissenschaftliche Fragestellungen des Moduls "Schwangere und Stillende" | 30 |
|---|---|---|
| 10.2 | Teilnehmerinnen am Modul "Schwangere und Stillende" | 30 |
| 10.3 | Untersuchungsproramm des Moduls "Schwangere und Stillende" | 31 |
| 11. Mo | dul "Kids & Family" | 32 |
| 11.1 | Wissenschaftliche Fragestellungen des Moduls "Kids & Family" | 32 |
| 11.2 | Teilnehmende am Modul "Kids & Family" | 33 |
| 11.3 | Untersuchungsprogramm des Moduls "Kids & Family" | 33 |
| 12. Qua | alitätsmanagement | 35 |
| 13. Dat | tenschutz, Informationssicherheit und Datenmanagement | 35 |
| 13.1 | Arten personenbezogener Daten | 36 |
| 13.2 | Übergeordnete Prinzipien | 36 |
| 13.3 | Organisationsstruktur aus Sicht des Datenmanagements | 37 |
| 13.4 | Pseudonymisierung | 39 |
| 13.5 | Aufbewahrungsfristen | 39 |
| 13.6 | Datennutzung, Datenweitergabe und Datenempfänger | 40 |
| 14. Eth | ik | 40 |
| 14.1 | Ethische Grundsätze | 40 |
| 14.2 | Aufklärung und Einwilligung | 41 |
| 14.3 | Widerrufsrecht | 43 |
| 14.4 | Risiken bei Befragungen und Untersuchungen | 44 |
| 14.5 | Möglicher Nutzen für die Teilnehmenden | 45 |
| 14.6 | Versicherung für die Teilnehmenden und Aufwandsentschädigung | 45 |
| 15. Wis | ssenschaftlicher Beirat | 45 |
| Referen | zen | 47 |
| Anhang | | 52 |

#### 1. Hintergrund

Das Interesse an einer fleischlosen Ernährung steigt in Deutschland seit einigen Jahren stetig an. Basierend auf Marktforschungsdaten kann man derzeit von ca. sechs Millionen Vegetariern und knapp einer Million Veganern in Deutschland ausgehen [1, 2]. Laut einer Umfrage, die vom Bundesministerium für Ernährung und Landwirtschaft (BMEL) beauftragt wurde, sank der Anteil der Personen, die angaben, täglich Fleisch zu verzehren, seit 2015 von 34 % auf 26 % [3].

Frühere Studien beschreiben positive Effekte einer vegetarischen und veganen Ernährung insbesondere auf die Entwicklung einer Adipositas und eines Typ-2-Diabetes [4]. Aus einer systematischen Übersichtsarbeit geht hervor, dass eine vegetarische Ernährung mit einem geringeren Risiko für ischämische Herzkrankheiten und Krebs assoziiert ist (basierend auf fünf bzw. zwei Studien) [5]. Auch eine vegane Ernährung geht demnach mit einem geringeren Krebsrisiko einher (basierend auf zwei Studien). Diese Übersichtsarbeit beruht überwiegend auf Kohortenstudien mit Rekrutierung in den 1980er und 1990er Jahren. Daten der European Prospective Investigation into Cancer and Nutrition (EPIC)-Studie aus Oxford (Basiserhebung von 1993 bis 2001) zeigen nach 18 Jahren Beobachtungszeit für Pescetarier (Personen, die kein Fleisch, jedoch Fisch verzehren) ein geringeres Risiko, einen Diabetes Typ 2 zu entwickeln als für Mischköstler oder Vegetarier [6]. Die in früheren Studien untersuchten Expositionen sind aufgrund des damaligen Lebensmittelangebots jedoch nur bedingt mit heutigen pflanzenbasierten Ernährungsweisen vergleichbar. Der Verzicht auf tierische Lebensmittel kann zudem mit einer unzureichenden Nährstoffzufuhr einhergehen [7]. Auch nimmt das Angebot an veganen Lebensmitteln und Fleischalternativprodukten in den letzten Jahren stetig zu. Dabei handelt es sich teilweise um hochverarbeitete bzw. zucker-, fett- oder salzreiche Lebensmittel, deren Verzehr laut einer aktuellen Studie bei Veganern einen Anteil von 39 % der Gesamtenergiezufuhr ausmachen kann [8]. Somit kann der Verzicht auf Fleisch oder jegliche tierische Produkte nicht mit einer gesunden Ernährungsweise gleichgesetzt werden. Auswertungen der Nationalen Verzehrsstudie II zeigen in Bezug Umweltkontaminanten tendenziell geringere Aufnahmen an Dioxinen und dioxinähnlichen polychlorierten Biphenylen bei vegetarischer Ernährung im Vergleich zur Allgemeinbevölkerung, jedoch tendenziell höhere Aufnahmen an Cadmium und Blei [9-11]. Für eine höhere Cadmiumaufnahme bei Vegetariern und Veganern verglichen mit Mischköstlern spricht auch der Vergleich der Cadmiumgehalte im Blut in einer tschechischen Studie [12]. Ergebnisse der EPIC-Oxford-Studie deuten nach 18 Jahren Nachbeobachtung darauf hin, dass Vegetarier ein höheres Schlaganfallrisiko als Mischköstler haben [13]. Zwei Meta-Analysen berichten eine geringere Knochendichte und ein höheres Frakturrisiko bei Veganern verglichen mit Mischköstlern [14]. Auch scheint das Risiko des Auftretens einer Depression bei Personen

mit veganer oder vegetarischer Ernährungsweise laut eines kürzlich publizierten systematischen Reviews mit Meta-Analyse erhöht zu sein [15].

Trotz des wachsenden Interesses an pflanzenbasierter Ernährung und der zunehmenden Diskussion über deren Risiken und Vorteile sind aktuelle Studien, die den damit verbundenen Gesundheitsstatus und insbesondere langfristige Gesundheitseffekte untersuchen, rar [16]. In Deutschland durchgeführte Studien mit erwachsenen Veganern und Vegetariern stammen überwiegend aus den 1980er und 1990er Jahren [17, 18] und repräsentieren damit keine pflanzenbasierte Ernährung aus heutiger Sicht. Zum Ernährungsstatus von Erwachsenen mit pflanzenbasierter Ernährung sind lediglich zwei aktuelle Studien aus Deutschland verfügbar: die Nutritional Evaluation (NuEva)-Study aus Jena, mit 58 Veganern, 65 Vegetariern, 70 Flexitariern (Personen, die nur gelegentlich Fleisch verzehren) und 65 Mischköstlern [19] und die Risks and Benefits of a Vegan Diet (RBVD)-Study des Bundesinstituts für Risikobewertung (BfR) mit 36 Veganern und 36 Mischköstlern [20]. Beide Studien lassen jedoch aufgrund ihres Querschnittsdesigns und der geringen Teilnehmendenzahlen keine Rückschlüsse auf längerfristige oder kausale Effekte pflanzenbasierter Ernährungsformen zu.

Das Nationale Ernährungsmonitoring generiert repräsentative Daten zu Lebensmittelverzehr, Nährstoffzufuhr, Nährstoffstatus und weiteren Aspekten des Ernährungsverhaltens der deutschen Bevölkerung im Alter von 18 bis 80 Jahren [21]. Es wird zurzeit mit kontinuierlichen Erhebungen neu konzipiert. Aufgrund der geplanten Teilnehmendenzahlen von 2.500 je Erhebung werden Auswertungen für kleine Subgruppen wie Personen mit besonderen Ernährungsweisen jedoch nicht möglich sein. Die Daten des Ernährungsmonitorings dienen zudem nur der Beschreibung der Ernährungssituation der Bevölkerung.

Auch für die Schwangerschaft und Stillzeit liegen kaum aktuelle Daten aus Deutschland zu Vorteilen oder Risiken einer pflanzenbasierten Ernährung vor. Bei einer veganen oder vegetarischen Ernährung während der Schwangerschaft scheint das Risiko einer exzessiven Gewichtszunahme oder eines Gestationsdiabetes im Vergleich zu einer Mischkost potenziell geringer zu sein. Dagegen kann das Risiko für ein erniedrigtes Geburtsgewicht des Kindes höher sein [22, 23]. Hinsichtlich einer Frühgeburtlichkeit scheint kein Unterschied oder ein eher geringeres Risiko zu bestehen [24, 25].

Für Kinder und Jugendliche fehlen ebenfalls Daten zum Nährstoffstatus und gesundheitlichen Folgen pflanzenbasierter Ernährungsweisen, trotz deren zunehmender Beliebtheit in dieser Altersgruppe [26, 27]. Die Ergebnisse der wenigen vorhandenen nationalen und internationalen Studien überwiegend im Querschnittsdesign sind inkonsistent. Sie deuten sowohl auf potentiell positive (vor allem auf metabolische Parameter) als auch negative (unter anderem auf Wachstum und Knochenmineralisierung) gesundheitliche Effekte hin [28-34]. Daten der Vegetarian and Vegan Children and Youth (VeChi) Study, einer Querschnittsstudie aus Deutschland, zeigen altersgemäße anthropometrische Maße und unterschiedliche

Zufuhrmengen von Makronährstoffen bei ähnlicher Gesamtenergieaufnahme [35]. Die vorhandene Datenlage erlaubt keine Schlussfolgerungen auf gesundheitliche Langzeitfolgen einer im Kindesalter beginnenden und über längere Zeit praktizierten veganen oder vegetarischen Ernährung. Darüber hinaus fehlen Daten zu Zusammenhängen zwischen pflanzenbasierten Ernährungsformen der Eltern und der Ernährung ihrer Kinder. Obwohl die Familie und familiäre Essgewohnheiten vor allem bei jüngeren Kindern das Essverhalten wesentlich beeinflussen können [36-39], wurden diese Faktoren im Kontext einer veganen oder vegetarischen Ernährung bisher kaum untersucht. In Deutschland wird das Abendessen von 96 % der 6- bis 11-Jährigen und 79 % der 12- bis 17-Jährigen als gemeinsame Familienmahlzeit eingenommen [40]. Diese Zahlen verdeutlichen, dass Familienmahlzeiten das Ernährungsverhalten von Kindern über soziale und psychologische Mechanismen entscheidend prägen können.

Eine besondere Herausforderung für Studien zu pflanzenbasierter Ernährung ist die umfassende und valide Erhebung des Verzehrs veganer und vegetarischer Lebensmittel. Diese Lebensmittel sind in den verfügbaren Datenquellen nicht ausreichend abgebildet. Groß angelegte epidemiologische Studien wie die NAKO Gesundheitsstudie [41] erlauben daher derzeit keine eingehende gesundheitliche Bewertung pflanzenbasierter Ernährungsweisen. Der Anteil an Vegetariern und insbesondere Veganern ist zudem in Studien an der Allgemeinbevölkerung wie der NAKO und laufenden internationalen Studien (wie NutriNet Santé [42] oder UK Biobank [43]) zu gering, um gesundheitsbezogene Aussagen statistisch absichern zu können. Des Weiteren fehlen Daten zu den Hintergründen und der Dauer pflanzenbasierter Ernährungsweisen. Auch Biobanken und Biomarkermessungen bestehender epidemiologischer Studien sind nicht auf konkrete Fragestellungen zu pflanzenbasierter Ernährung ausgerichtet.

Aufgrund des Mangels an Daten und Forschungsressourcen sind Ernährungsempfehlungen für vegetarisch und vor allem vegan lebende Menschen derzeit nicht ausreichend evidenzbasiert.

Ernährungsweisen wirken sich auf Prozesse im gesamten Ernährungssystem aus und spielen eine Schlüsselrolle für eine nachhaltige und zukunftsfähige Entwicklung [44-46]. Es ist daher von hoher Relevanz, neben den gesundheitlichen Effekten einer pflanzenbasierten Ernährung auch soziale, ökologische und ökonomische Auswirkungen zu untersuchen. Bereits seit vielen Jahren fordern zahlreiche Stimmen aus Wissenschaft, Zivilgesellschaft und Politik auf nationaler und internationaler Ebene eine grundlegende Umgestaltung der Ernährungssysteme und eine Transformation zu mehr Nachhaltigkeit, die Lebensmittelversorgung der wachsenden Bevölkerung langfristig zu sichern [46-50]. Eine nachhaltige Ernährung sollte auf Bevölkerungsebene gesundheitsfördernd und erschwinglich sein sowie sich entlang der Wertschöpfungskette von Produktion über Verarbeitung und Handel bis hin zum Verzehr an Umweltschutz, Tierwohl und sozialen Standards ausrichten [50]. Die Autoren des Berichts der EAT-Lancet Kommission [44] empfehlen westlichen Industrienationen, ihre Ernährungsweise zu ändern und beispielsweise den Konsum von Obst und Gemüse zu verdoppeln sowie den Fleisch- und Zuckerkonsum zu halbieren. In der eingangs erwähnten Umfrage im Auftrag des BMEL [3] gaben 41 % der Befragten, die vegetarische oder vegane Alternativen zu tierischen Produkten gekauft hatten, Klimaschutzgründe für ihre Entscheidung an.

Der bisherige Wissensstand legt nahe, dass der Verzehr pflanzlicher Lebensmittel als Alternative zum Verzehr tierischer Lebensmittel vorteilhaft sein kann, insbesondere hinsichtlich gesundheitlicher und ökologischer Folgen [51-55]. Allerdings lässt sich diese Frage aufgrund der zunehmenden Lebensmittelvielfalt (z. B. bei hoch verarbeiteten Fleischalternativprodukten), heterogener Produktionsweisen und Bezugsmöglichkeiten sowie der Komplexität ernährungsbezogener Handlungen nicht pauschal beantworten. Hinzu kommt, dass zu den sozialen Folgen [50], aber auch den ökonomischen Auswirkungen der Ernährung bisher keine ausreichenden und kaum differenzierte Erkenntnisse vorliegen, die Aussagen zu potenziellen Vorteilen bestimmter Ernährungsweisen zulassen. Es fehlt zudem eine umfassende Nachhaltigkeitsanalyse von Ernährungsweisen, die die Dimensionen Gesundheit, Umwelt, Gesellschaft, und Wirtschaft in eine Gesamtbetrachtung integriert.

Aus dem vorgestellten Forschungsstand leiten sich die wissenschaftlichen Ziele der Studie ab, die im Folgenden beschrieben werden.

#### 2. Wissenschaftliche Ziele der COPLANT-Studie

Die Kohortenstudie zu pflanzenbasierter Ernährung "COhort on PLANT-based Diets (COPLANT) Study" zielt darauf ab, langfristige gesundheitliche Vorteile und mögliche Gesundheitsrisiken sowie soziale, ökologische und ökonomische Auswirkungen verschiedener pflanzenbasierter Ernährungsformen im Vergleich zu einer Mischkost zu untersuchen.

Die Studie soll wissenschaftliche Grundlagen für eine Überprüfung und mögliche Änderungen der Empfehlungen für eine gesunde Ernährung im deutschsprachigen Raum bereitstellen. Die Ergebnisse der Studie können die gesundheitliche Bewertung ernährungsassoziierter Risikofaktoren erheblich verbessern sowie Erkenntnisse zu einem breiten Spektrum möglicher Auswirkungen befördern. Sie sollen allen interessierten Gruppen als wichtige Entscheidungshilfe für gesundheitsbezogene und nachhaltigkeitsrelevante Maßnahmen dienen.

Mit dieser umfassenden Betrachtung bisher unzureichend charakterisierter Ernährungsweisen grenzt sich die Studie von laufenden epidemiologischen Studien in Deutschland deutlich ab.

Im Einzelnen werden die folgenden vier wissenschaftlichen Ziele verfolgt:

#### Ziel 1: Umfassende Erhebung der Ernährungsweise

- Umfassende Charakterisierung des Lebensmittelverzehrs und der Nährstoffzufuhr von Personen mit pflanzenbasierten Ernährungsweisen
- Untersuchung von Unterschieden in Lebensmittelverzehr und Nährstoffzufuhr zwischen verschiedenen Ernährungsweisen unter Berücksichtigung weiterer Lebensstilfaktoren
- Charakterisierung und Vergleich der externen und internen Aufnahme von Nährstoffen und Kontaminanten für Personen mit pflanzenbasierten Ernährungsweisen
- Untersuchung der Belastung mit Kontaminanten in Abhängigkeit von der Ernährungsweise und anderen Lebensstilfaktoren
- Risiko-Nutzen-Abwägungen für pflanzenbasierte Ernährungsweisen unter Berücksichtigung der Nährstoffversorgung und der Aufnahme unerwünschter Stoffe
- Einsatz und Weiterentwicklung digitaler Instrumente zur Erhebung des Lebensmittelverzehrs einschließlich der Erweiterung dafür verfügbarer Datenbanken
- Weiterentwicklung ernährungsassoziierter Biomarker

## Ziel 2: Analyse von Zusammenhängen der Ernährungsweise mit dem Gesundheitszustand und dem Auftreten chronischer Erkrankungen

Im Querschnitt (perspektivisch auch im Längsschnitt) sollen Assoziationen pflanzenbasierter Ernährungsweisen mit folgenden Merkmalen untersucht werden:

- Sozioökonomischer Status (Bildung, Beruf, Einkommen)
- Lebensstilfaktoren (z. B. körperliche Aktivität, Rauchen, Schlafverhalten)
- Körpermaße (Gewicht, Taillen- und Hüftumfang) und Körperzusammensetzung (Anteil und Verteilung von Körperfett und Muskelmasse)
- Risikofaktoren f
   ür kardiovaskul
   äre Erkrankungen (z. B. Blutlipide)
- (chronische) Entzündung
- Knochengesundheit
- Schilddrüsenfunktion
- Intestinales Mikrobiom
- Metabolom
- Epigenetik
- Mentale Gesundheit

Im Längsschnitt sollen folgende Themen untersucht werden (auch im Zusammenschluss mit internationalen Studien):

- Ernährungsweise und intermediäre Marker
- Ernährungsweise und Inzidenz chronischer Erkrankungen (darunter Typ 2 Diabetes, Herz-Kreislauf-Erkrankungen, Krebserkrankungen, Osteoporose, Depression)
- Veränderungen pflanzenbasierter Ernährungsweisen im Lebenszyklus

#### Ziel 3: Überprüfung bestehender Ernährungsempfehlungen

- Berücksichtigung der Bedeutung neuer, verarbeiteter Produkte auf Pflanzenbasis
- Ableitung von Empfehlungen vor allem für vegetarisch und vegan lebende Menschen in enger Zusammenarbeit mit Fachgesellschaften und Vertretern der vegetarischen und veganen "Community"
- Aufbau eines Netzwerks aus dem Konsortium der Antragsteller für Wissenstransfer und Nutzen-Risiko-Kommunikation mit großer Reichweite

#### Ziel 4: Analyse der Nachhaltigkeit verschiedener Ernährungsweisen

- Charakterisierung der verschiedenen Ernährungsweisen hinsichtlich ihrer sozialen (einschließlich ethischen und kulturellen), ökologischen und ökonomischen Auswirkungen, unter Berücksichtigung ausgewählter Aspekte bei Beschaffung, Zubereitung, Verzehr und Nachbereitung von Lebensmitteln
- Entwicklung eines Instruments zum Vergleich der Ernährungsweisen hinsichtlich deren Nachhaltigkeit bezogen auf die Dimensionen Gesundheit, Umwelt, Gesellschaft und Wirtschaft
- Untersuchung von Determinanten für nachhaltiges Ernährungsverhalten (z. B. Motivationen, Werthaltungen, Hemmnisse)
- Ableitung von Handlungsbedarfen und -optionen für eine Veränderung des Ernährungsverhaltens hin zu mehr Nachhaltigkeit
- Untersuchung von Veränderungen in der Nachhaltigkeit von Ernährungsweisen über die Zeit sowie von langfristigen Gesundheitsauswirkungen nachhaltiger pflanzenbasierter Ernährungsweisen

#### 3. Studienzentren, assoziierte Partner und Verantwortlichkeiten

Die COPLANT-Studie soll an acht Standorten durchgeführt werden. Die nachfolgenden Institutionen, die auch die Rekrutierung von Studienteilnehmenden in einem Studienzentrum beabsichtigen, sind aufgrund ihrer wissenschaftlichen Expertise im Hinblick auf die Fragestellungen der Studie und ihrer praktischen Erfahrungen mit Kohortenstudien an einer gemeinsamen Durchführung der Studie interessiert. Die Studienzentren verteilen sich in Deutschland auf folgende Forschungseinrichtungen: Bundesinstitut für Risikobewertung (BfR) Berlin, Max Rubner-Institut (MRI) Karlsruhe, Rheinische Friedrich-Wilhelms-Universität Bonn, Friedrich-Schiller-Universität Jena, Universität Heidelberg, Universität Regensburg und Forschungsinstitut für pflanzenbasierte Ernährung Gießen. In Österreich richtet die Universität Wien ein Studienzentrum ein. Vertreterinnen und Vertreter aller Studienzentren nahmen an Planungstreffen, die dem Studienstart vorausgingen, teil.

Das BfR übernimmt zentrale Organisationsaufgaben und das Datenmanagement. Die Universität Bonn stellt in Zusammenarbeit mit dem BfR die NutriDiary-App für die Ernährungserhebung bereit. Das Johann Heinrich von Thünen-Institut ist assoziierter Partner der COPLANT-Studie und leitet gemeinsam mit dem MRI das Teilprojekt Nachhaltigkeitsanalyse. Das Universitätsklinikum Jena übernimmt als assoziierter Partner zusammen mit dem BfR die Lagerung von Blut- und Urinproben für die Laufzeit der Rekrutierung der Studienteilnehmenden. Das MRI ist für das Lagern und Versenden der Stuhlproben verantwortlich.

Zudem bestehen ein intensiver Austausch zur Studienplanung mit Wissenschaftlerinnen und Wissenschaftlern des Instituts für Epidemiologie, Biostatistik und Prävention der Universität Zürich sowie der Fachhochschule Bern (Schweiz). Ziel ist es, bei eigener Finanzierung eines Studienzentrums das Design der COPLANT-Studie weitestgehend zu übernehmen, so dass zukünftig gemeinsame Auswertungen der erhobenen Daten möglich sein werden.



Abbildung 1 Beteiligte Studienzentren

Jedes Studienzentrum besitzt eine Zentrumsleitung (Tabelle 1). Die Abläufe im Studienzentrum und der Einsatz des Personals werden im jeweiligen Studienzentrum eigenständig koordiniert. Insbesondere soll gewährleistet werden, dass die Teilnehmenden durch geschultes Personal aufgeklärt werden, bei medizinischen Notfällen eine ärztliche Rufbereitschaft sichergestellt ist, der Datenschutz nach Datenschutz-Grundverordnung (DSGVO) und die Informationssicherheit bei der Datenerhebung eingehalten werden.

Tabelle 1 Beteiligte Studienzentren und deren Leitung

| Studienzentrum | Studienzentrumsleitung |
|---|---|
| Bundesinstitut für Risikobewertung,<br>Berlin | Prof. Dr. Cornelia Weikert Fachgruppe Risiken besonderer Bevölkerungsgruppen und Humanstudien Max-Dohrn-Straße 8-10 10589 Berlin |
| Max Rubner-Institut, Karlsruhe | Dr. Benedikt Merz Bundesforschungsinstitut für Ernährung und Lebensmittel Institut für Physiologie und Biochemie der Ernährung Haid-und-Neu-Straße 9 76131 Karlsruhe |
| Rheinische Friedrich-Wilhelms-Universität Bonn | Prof. Dr. Ute Nöthlings<br>Institut für Ernährungs- und Lebensmittelwissenschaften<br>Friedrich-Hirzebruch-Allee 7<br>53115 Bonn |
| Forschungsinstitut für pflanzenbasierte Ernährung, Gießen | Dr. Markus Keller<br>Forschungsinstitut für pflanzenbasierte Ernährung (IFPE)<br>gGmbH<br>Am Lohacker 2<br>35444 Biebertal/Gießen |
| Friedrich-Schiller-Universität Jena | Dr. Christine Dawczynski<br>Institut für Ernährungswissenschaften<br>Dornburger Straße 29<br>07743 Jena |
| Universität Regensburg | Prof. Dr. Dr. Michael Leitzmann Institut für Epidemiologie und Präventivmedizin Universitätsklinikum Regensburg Franz-Josef-Strauß-Allee 11 93053 Regensburg |
| Universität Heidelberg | JunProf. Dr. Ina Danquah<br>Institut für Global Health<br>Im Neuenheimer Feld 130.3<br>69120 Heidelberg |
| Universität Wien | Prof. Dr. Maria Wakolbinger Prof. Dr. Tilman Kühn Zentrum für Public Health, Public Health Nutrition; Medizinische Universität Wien Kinderspitalgasse 15/1 1090 Wien |

#### 4. Projektkoordination

Die Projektkoordination obliegt dem BfR und umfasst folgende Aufgaben:

- Koordination des Gesamtprojektes
- Zentrale Datenhaltung (Forschungsdatenbank und Treuhandstelle)

- Koordination des Qualit\u00e4tsmanagements, einschlie\u00dflich zentraler Schulungen und Zertifizierungen sowie Monitoring der Datenqualit\u00e4t
- Öffentlichkeitsarbeit

Insbesondere sind die Arbeiten der Projektpartner sachlich und zeitlich zu koordinieren. Die Projektkoordination bereitet die für die Arbeits- und Zeitplanung notwendigen Treffen der Studienzentren vor, lädt dazu mit einer angemessenen Frist unter Beifügung der Tagesordnung ein, führt den Vorsitz bei den Arbeitssitzungen, erstellt und versendet die Sitzungsprotokolle. Neben der lokalen Datensammlung in den einzelnen Studienzentren werden am BfR eine gemeinsame Datenbank und ein zentrales Datenmanagement aufgebaut und implementiert. Die Studienzentren werden die Studiendaten, wenn möglich gemeinsam, aber wenn notwendig auch von einzelnen Studienzentren auswerten. Entsprechende Vereinbarungen der Zusammenarbeit finden sich im Kooperationsvertrag, der Nutzungsordnung und der Publikationsordnung.

Alle Datenerhebungen der COPLANT-Studie unterliegen einem umfassenden Qualitätsmanagement (Kapitel 12). Grundlage der Qualitätssicherung der Untersuchungen, Befragungen und Probenverarbeitung sind die vor Studienbeginn erstellten standardisierten Arbeitsanweisungen (Standard Operating Procedures, SOPs). Das Studienpersonal wird vor Studienbeginn für alle Datenerhebungen theoretisch und praktisch geschult, supervisiert und zertifiziert.

#### 5. Studiendesign

#### 5.1 Studientyp

Es wird eine prospektive bevölkerungsbasierte Kohortenstudie mit ca. 6000 Frauen und Männern im Alter von 18 bis 69 Jahren aufgebaut.

In Abhängigkeit von der seit mindestens einem Jahr praktizierten Ernährungsweise werden die Studienteilnehmenden einer der folgenden vier Gruppen (Studienexposition) zugeordnet:

#### Veganer

kein Verzehr tierischer Produkte (weniger als eine Ausnahme monatlich)

#### Vegetarier

- kein Verzehr von Fleisch und Fisch (weniger als eine Ausnahme monatlich)
- Verzehr von Eiern und/oder Milchprodukten (mindestens einmal monatlich)

#### **Pescetarier**

- kein Verzehr von Fleisch (weniger als eine Ausnahme monatlich)
- Verzehr von Fisch (mindestens einmal monatlich)
- Verzehr von Eiern oder Milchprodukten möglich

#### Mischköstler (Omnivore) – Gruppe der Nicht-Exponierten bzw. Kontrollgruppe

- Verzehr von Fleisch oder Wurst (mindestens einmal monatlich).

Die Basiserhebung wird sich über ca. drei Jahre erstrecken (Abbildung 2). Sie umfasst die Erhebung der Ernährungsweise und eine umfangreiche Phänotypisierung von Veganern, Vegetariern, Pescetariern und Omnivoren.

Bei der geplanten Nachbeobachtung werden die Studienteilnehmenden in regelmäßigen Abständen schriftlich kontaktiert, um Veränderungen der Ernährungsweise, des Lebensstiles und des Gesundheitsstatus mithilfe von Fragebögen zu erfassen. Bei erfolgreicher Einwerbung von Drittmitteln wird nach fünf bis zehn Jahren erneut ins Studienzentrum eingeladen. Zusätzlich wird eine passive Nachbeobachtung mittels Sekundärdaten angestrebt.



Abbildung 2 Design der COPLANT-Studie

#### 5.2 Ein- und Ausschlusskriterien

In die Studie eingeschlossen werden interessierte Personen, die

- zum Zeitpunkt der Rekrutierung zwischen 18 und 69 Jahren alt sind
- ihrer aktuellen Ernährungsweise seit mindestens einem Jahr folgen
- krankenversichert sind
- zur Blutentnahme und zum Ausfüllen von Fragebögen bereit sind
- nur an den Standorten Regensburg, Heidelberg, Bonn und Wien: zum Zeitpunkt der Rekrutierung weder schwanger sind noch stillen (Kapitel 10)
- die Anforderungen der Studie sprachlich und inhaltlich verstehen und nach Aufklärung zur Einwilligung in die Studienteilnahme fähig sind
- ihre Einwilligung zur Teilnahme an der COPLANT-Studie gegeben haben.

Aus der Studie ausgeschlossen werden Studienteilnehmende,

• die nicht mehr kontaktiert werden können

die ihre Zustimmung zur Teilnahme an der Studie widerrufen.

#### 5.3 Rekrutierung der Studienteilnehmenden

Die Studienteilnehmenden werden als so genanntes "Convenience Sample", z. B. über Aushänge sowie lokale und soziale Medien, rekrutiert. An einer Teilnahme interessierte Personen können sich per Post, per E-Mail oder telefonisch in einem der acht Studienzentren melden. Nachdem sich Studieninteressenten im Studienzentrum gemeldet haben, werden sie telefonisch kontaktiert. Dabei wird anhand eines Kurzfragebogens geprüft und entschieden, ob die Person die Einschlusskriterien der Studie erfüllt. Bei Eignung für die Studie wird der erste Termin im Studienzentrum vereinbart. Informationen zur Studie und die Einwilligungserklärung werden nachfolgend per E-Mail versandt. In der Studieninformation erhalten die Studieninteressenten Informationen zu wichtigen Aspekten der Studie, wie Teilnahmebedingungen, Untersuchungsprogramm, potenzielle Risiken (z. B. durch die Blutentnahme), Mitteilung von persönlichen Untersuchungsergebnissen, Probenaufbewahrung, beabsichtigte und mögliche weitere Datenanalysen (einschließlich klinisch-chemische, molekulare und genetische Analysen), Freiwilligkeit, Recht auf Widerruf, Vertraulichkeit, Datenschutz und Ansprechpersonen. Bei Unklarheiten können die Studieninteressenten bei ihrem Erstbesuch im Studienzentrum, per E-Mail oder während der Telefonsprechzeiten nachfragen.

Der Kurzfragebogen im Rahmen des telefonischen Erstkontakts weist die Studieninteressenten auch einer der vier Ernährungsgruppen zu. Da eine pflanzenbasierte Ernährung vor allem bei jüngeren Frauen anzutreffen ist, werden die Mitglieder der vier Ernährungsgruppen stratifiziert nach Geschlecht und Alter rekrutiert, um Aussagen für die gesamte Bevölkerung treffen zu können. Es wird in vier Altersgruppen (18 bis 29, 30 bis 39, 40 bis 49 und 50 bis 69 Jahre) rekrutiert. Bei zu erwartenden Schwierigkeiten bei der Rekrutierung älterer Personen wird eine ungleiche Besetzung der Strata zugelassen. Hinsichtlich der Geschlechtsverteilung werden gleiche Anteile von Frauen und Männern angestrebt, wobei ein Frauen-Anteil von bis zu 60 % akzeptiert wird.

Um die Teilnehmenden an COPLANT in allen Studienzentren nach einheitlichem Vorgehen zu rekrutieren, müssen die Kontaktaufnahme standardisiert erfolgen und das Vorgehen transparent dokumentiert werden. Für die Organisation und Dokumentation der Arbeitsabläufe bei der Rekrutierung wird in allen Zentren das **web**basierte **Mo**dulare Steuerungs- und **D**okumentationss**ys**tem (webMODYS) [56] verwendet. Es automatisiert Standardaktivitäten, wie das Generieren von E-Mails an Studienteilnehmende und das Zuordnen von Terminen. WebMODYS stellt verschiedene Informationen über den Fortgang der Studie, darunter Auszählungen zur Beteiligung und die Erfassung von Gründen der Nichtteilnahme, zur Verfügung. Die erhobenen Daten können direkt verwendet werden, z. B. um Statistiken zu erstellen.

#### Einfluss der Rekrutierung auf die Validität der Studienergebnisse

Die Rekrutierung von Interessenten an den Forschungsfragen der COPLANT-Studie wird mit einer Anreicherung gesundheitsbewusster Personen gegenüber der deutschen Allgemeinbevölkerung einhergehen. Als Konsequenz ist mit einer Überschätzung der Prävalenz gesundheitsfördernder Verhaltensweisen und einer Unterschätzung des Vorkommens gesundheitsschädigenden Verhaltens sowie dessen Folgen in COPLANT gegenüber der Zielbevölkerung zu rechnen. Unter der Annahme, dass omnivore Studienteilnehmende weniger und qualitativ hochwertigeres Fleisch verzehren als Omnivore in der Allgemeinbevölkerung, dürften zudem die gesundheitlichen Effekte pflanzenbasierter Ernährungsweisen in COPLANT unterschätzt werden.

Eine Rekrutierung über Einwohnermeldeämter mit dem Ziel, eine bevölkerungsrepräsentative Stichprobe zu erhalten, ist für die Fragestellungen von COPLANT jedoch nicht zielführend. Um 1600 Veganer in die Studie aufnehmen zu können, müssten aufgrund der geringen Prävalenz der veganen Ernährungsweise von 1 % [2] bei einer erwarteten Beteiligung von 20 % [41] insgesamt 1600\*100\*5 = 800.000 Personen kontaktiert werden. Die geringe erwartete Beteiligung weist zudem darauf hin, dass auch die Rekrutierung über Einwohnermeldeämter mit einer Selektion gesünderer Studienteilnehmender verbunden ist [41, 57].

#### 5.4 Zeitplan

Die Vorbereitungen der Studie, wie Finalisierung des Studienprotokolls, Klärung der Finanzierung, Entwicklung von Fragebögen, Aufbau der Logistik und eines Qualitätsmanagementsystems, begannen im 4. Quartal 2021. Das Ernährungserhebungsinstrument NutriDiary-App ist seit Januar 2023 für die Studie einsatzfähig. Ab Ende des 2. Quartals 2023 führen alle Studienzentren einen Prätest mit jeweils zwei Personen und ab Dezember 2023 eine Pilotstudie mit jeweils zehn Teilnehmenden durch (Abbildung 3). Nachdem mindestens vier Studienzentren die Pilotstudie absolviert haben, das Studienprotokoll auf Machbarkeit überprüft und bei Bedarf angepasst wurde, soll ab Anfang 2024 bis 2026 für die Hauptstudie rekrutiert werden. Bei erfolgreicher Einwerbung von Drittmitteln werden die Studienteilnehmenden alle drei bis fünf Jahre schriftlich zu ihrem Gesundheitsstatus nachbefragt sowie alle fünf bis zehn Jahre erneut ins Studienzentrum eingeladen.



Abbildung 3 Zeitplan der COPLANT-Studie

FUP = Follow-up

#### 6. Basiserhebung

#### 6.1 Ablauf der Basiserhebung

Alle Studienteilnehmenden durchlaufen bei zwei Besuchen im lokalen Studienzentrum ein Untersuchungsprogramm und füllen einen Fragebogen computergestützt aus (Abbildung 4). Von jedem Teilnehmenden werden darüber hinaus Blut-, Urin- und Stuhlproben gewonnen. Alle Datenerhebungen werden standardisiert nach einheitlichen SOPs von geschultem Personal durchgeführt.

Beim ersten Besuch im Studienzentrum werden die Studieninteressenten in einem persönlichen Gespräch über die Studie aufgeklärt. Sie unterschreiben die Einwilligungserklärung und werden damit zu Studienteilnehmenden. Sie erhalten die Studienmaterialien (Küchenwaage, Sammelbehälter für Urin und Stuhl, Kühltasche, Akzelerometer) und Anleitungen zu deren Handhabung. Die Teilnehmenden werden in die Ernährungserhebung mittels NutriDiary-App und in die Protokollierung ihrer Lebensmittelabfälle eingeführt. Sie füllen den Großteil des Fragebogens (Module Soziodemografie, Ernährung, Verhalten im Alltag Teil 1, Gesundheit, Tabelle 2) aus und werden über die Möglichkeit, an einem vertiefenden Interview zu persönlichen Perspektiven auf Ernährung teilzunehmen, informiert (Kapitel 9). Bei Interesse unterschreiben die Teilnehmenden eine separate Einwilligungserklärung zur späteren Rekontaktierung. Zudem werden Blutdruck, Puls und Handgreifkraft bestimmt. Der erste Besuch dauert zwei bis drei Stunden.



Abbildung 4 Programm der Basiserhebung der COPLANT-Studie

Zwischen dem ersten und zweiten Besuch im Studienzentrum führen die Teilnehmenden drei eintägige Wiege-Ernährungsprotokolle mittels NutriDiary-App, tragen über bis zu sieben Tage einen Aktivitätssensor, füllen das Modul Lebensstil des Fragebogens aus und protokollieren während der drei Tage vor dem zweiten Besuchstermin ihre Lebensmittelabfälle.

Der zweite Besuch findet zwei bis vier Wochen nach dem ersten Besuch statt. Die Teilnehmenden erscheinen nüchtern zum Termin für eine Blutentnahme. Sie geben einen Sammelurin vom Vortag und eine am Morgen des Besuchstages entnommene Stuhlprobe ab. Die Teilnehmenden füllen einen Verzehrshäufigkeitsfragebogen (FFQ), einen Fragebogen zu den Lebensmittelabfällen sowie das Modul Verhalten im Alltag Teil 2 des Hauptfragebogens (Tabelle 2) am PC aus. In einem computergestützten Interview wird die Einnahme von Arzneimitteln und Nahrungsergänzungsmitteln erhoben. Blutdruck, Körpermaße und Körperzusammensetzung sowie die Knochengesundheit werden bestimmt. Optional kann jedes Studienzentrum noch weitere Untersuchungen (z. B. Sonographie der Schilddrüse) durchführen. Der zweite Besuch dauert drei bis vier Stunden.

In Berlin werden die Teilnehmenden vier bis acht Wochen nach dem zweiten Besuch zu einem dritten Besuch in das Studienzentrum eingeladen. Am Vortag führen sie ein viertes Wiege-Ernährungsprotokoll und sammeln ihren Urin. Am Morgen des Besuchstages nehmen sie erneut eine Stuhlprobe. Im Studienzentrum wird nochmals Blut entnommen. Die Teilnehmenden füllen einen zweiten FFQ sowie einen Fragebogen zur Ernährungskompetenz am PC aus.

#### Nichtteilnahme an der Basiserhebung

Studienteilnehmende, die im Verlauf der Basiserhebung nicht mehr kontaktiert werden können oder ihre Einwilligung zur Teilnahme an der Studie widerrufen, werden von der weiteren Teilnahme an COPLANT ausgeschlossen. Personen, die die weitere Studienteilnahme temporär ablehnen, z. B. aus zeitlichen oder gesundheitlichen Gründen, können dagegen im Studienverlauf erneut kontaktiert werden. Die Gründe für ein Ausscheiden aus der Studie werden in der Rekrutierungs-Software webMODYS dokumentiert.

#### 6.2 Erhebung der Ernährungsweise

Mit pflanzenbasierten Ernährungsweisen als Studienexposition ist die Erhebung von Ernährungsdaten ein Hauptinhalt der COPLANT-Studie. Mit der umfassenden Erhebung insbesondere veganer und vegetarischer Ernährungsweisen soll die Aufnahme potentiell gesundheitsfördernder oder -schädigender Substanzen bei diesen Ernährungsformen geschätzt werden. Für die Erhebung der Ernährung werden mehrere Instrumente eingesetzt (Abbildung 5):

- mindestens vier eintägige Wiegeprotokolle, die mithilfe einer Smartphone-basierten
   App geführt werden
- ein Verzehrshäufigkeitsfragebogen (Food Frequency Questionnaire, FFQ) zur Ernährung in den letzten zwölf Monaten, der webbasiert ausgefüllt wird
- ein computergestütztes Interview zur Einnahme von Nahrungsergänzungsmitteln in den letzten vier Wochen vor dem zweiten Besuch im Studienzentrum.



**Abbildung 5** Ablauf der Ernährungserhebung in der COPLANT-Studie WT = Wochentag, WE = Wochenendtag, B = Besuch im Studienzentrum, P = eintägiges Wiegeprotokoll, FFQ = Verzehrshäufigkeitsfragebogen, NEM = Erhebung von Nahrungsergänzungsmitteln

#### Ernährungserhebung mittels Wiegeprotokoll

Mit mehreren Wiegeprotokollen wird der Lebensmittelverzehr jeweils über einen Tag erhoben. Das in COPLANT eingesetzte Wiegeprotokoll basiert auf etablierten Instrumenten der DO-NALD- und KiESEL-Studien [58, 59]. Es unterscheidet sich davon lediglich durch die Erfassung der Verzehrsinformation mit einer Smartphone-basierten App anstelle eines Papierprotokolls. Studien belegen, dass digitale Instrumente zur Verzehrserhebung hinsichtlich der Genauigkeit keine wesentlichen Nachteile gegenüber herkömmlichen Instrumenten aufweisen [60, 61].

Für akute und chronische Risikobewertungen empfiehlt die European Food Safety Authority (EFSA) mindestens zwei individuell erhobene Verzehrstage [62, 63]. Dagegen zeigen Studien

zur Extrapolation von Kurzzeit- auf Langzeitaufnahmen, dass insbesondere bei höherer intraindividueller Variabilität des Lebensmittelverzehrs oder der Nährstoff- bzw. Schadstoffaufnahme mehr als zwei Verzehrstage erhoben werden sollten [64, 65]. Die Teilnehmenden an
COPLANT sind aufgefordert, zwischen den beiden Studienzentrumsbesuchen drei Wiegeprotokolle zu führen, davon eines an einem Wochenendtag (Abbildung 5). Zwei aufeinanderfolgende Wiegeprotokolle sollen unmittelbar vor dem zweiten Besuch geführt werden, um einen
direkten Bezug zu den an diesem Tag erhobenen Biomarkern herstellen zu können.

Beim zweiten Besuch im Studienzentrum wird ein vierter Tag für ein Wiegeprotokoll vereinbart. Dabei ist zu berücksichtigen, dass mindestens zwei der vier Protokolltage auf einen Wochentag fallen. Das vierte Protokoll sollte möglichst vier Wochen nach dem dritten Protokoll geführt werden, aber spätestens acht Wochen danach abgeschlossen sein. An den Standorten, an denen die Teilnehmenden einen dritten Besuchstermin erhalten (BfR und MRI), sollte der vierte Protokolltag unmittelbar vor diesem Termin liegen, um einen Bezug des protokollierten Verzehrs zu den Blut- und Urinmarkern sicherstellen zu können.

Nach Abschluss der vier Pflichtprotokolle sind die Teilnehmenden gebeten, zusätzliche eintägige Wiegeprotokolle zu führen. Hierzu erhalten sie im Abstand von jeweils 90 Tagen per E-Mail insgesamt drei Aufforderungen.

#### NutriDiary – App für Wiege-Ernährungsprotokolle

Die Wiege-Ernährungsprotokolle werden mit der App NutriDiary [66] geführt. Die Teilnehmenden werden über eine Webseite (Researcher Webseite) von den Studienzentren verwaltet. Die Studienzentren erhalten für ihre Teilnehmenden Zugangskodes. Die Verknüpfung von personenbezogenen Merkmalen liegt damit ausschließlich im Studienzentrum vor.

Die Teilnehmenden werden beim ersten Besuch im Studienzentrum gebeten, die NutriDiary-App auf ihr Smartphone herunterzuladen (Abbildung 6). Sie erhalten außerdem individuelle Zugangsdaten, mit denen sie sich in die Anwendung einloggen können.



**Abbildung 6** NutriDiary App und QR-Codes zum Herunterladen von NutriDiary aus dem App Store (oben für IOS, unten für Android)

Am vereinbarten Protokolltag wiegen und protokollieren die Teilnehmenden alle verzehrten Lebensmittel und Getränke. Diese können in der in die App integrierten Nährstoffdatenbank LEBTAB gesucht werden. Für die Suche der Lebensmittel haben die Teilnehmenden zwei Möglichkeiten: die textbasierte Suche und die Suche über die Barcode-Scanfunktion. Bei der textbasierten Suche wird die Bezeichnung des Lebensmittels in das Suchfeld der Lebensmitteleingabe eingetragen. Datenbankeinträge, die diese Bezeichnung enthalten, werden als Liste angezeigt. Ist das gesuchte Lebensmittel dabei, kann es aus der Liste ausgewählt und mit der Eingabe der zusätzlich abgefragten Informationen fortgefahren werden. Alternativ kann der Barcode eines Produktes gescannt werden. Ist ein Lebensmittel mit diesem Barcode in der Datenbank vorhanden, wird seine Bezeichnung automatisch im Suchfeld der Lebensmitteleingabe angezeigt.

Ist ein Produkt noch nicht in der Datenbank hinterlegt, sind die Teilnehmenden aufgefordert, das Produkt zu fotografieren. Die Fotos (Barcode, Produktname/-marke, Zutatenliste, Nährwerttabelle) werden an einen Server geschickt, wo Algorithmen des maschinellen Lernens Informationen von den Produktverpackungen extrahieren. Anhand dessen werden eine Rezeptsimulation durchgeführt und entsprechende Nährstoffdaten für das Produkt in LEBTAB ergänzt. Auf diese Weise wird die Datenbank kontinuierlich erweitert. Von Teilnehmenden neu angelegte Produkte sind unmittelbar für die Suche verfügbar.

Für jedes Lebensmittel sind neben der Bezeichnung und der abgewogenen Menge das Datum, die Uhrzeit und der Ort des Verzehrs einzutragen sowie die Zubereitungsart aus einer Liste auszuwählen. Lebensmittelreste und die Art der Erzeugung (biologisch oder konventionell) sind ebenso zu protokollieren. Wurde ein Verzehrstag vollständig protokolliert, beenden die

Teilnehmenden das Wiegeprotokoll in der App. Auf der Researcher Webseite können die Studienzentren für ihre Teilnehmenden einsehen, ob bereits Lebensmittel protokolliert wurden oder ein Protokoll abgeschlossen wurde. Anhand der ebenfalls sichtbaren Anzahl protokollierter Items sind im Studienzentrum Rückfragen im Sinne einer ersten Qualitätskontrolle möglich. Die abgeschlossenen Protokolle werden an den NutriDiary-Server an der Universität Bonn gesendet, wo sie Mitarbeitende der Professur Ernährungsepidemiologie herunterladen können. Diese prüfen die Protokolle auf Plausibilität und übermitteln sie nach weiteren Verarbeitungsschritten zur Datenaufbereitung (Datenbereinigung, Kodierung, Lebensmittelgruppierungen usw.) an das zentrale Datenmanagementsystem REDCap.

Der Ablauf der Ernährungserhebung vom Anlegen der Benutzerkonten bis zum vollständig kodierten Ernährungsprotokoll ist im Anhang A1 dargestellt.

Die Wiegeprotokolle können auf Wunsch auch auf Papier geführt werden. Dafür erhalten die Teilnehmenden beim ersten Besuch im Studienzentrum entsprechende Vordrucke. Geschulte Mitarbeitende der Studienzentren geben die Papierprotokolle nachträglich in die NutriDiary-App ein. Die weitere Datenverarbeitung erfolgt wie oben beschrieben. Eine Kombination von App- und papierbasierter Protokollierung des Verzehrs ist nicht möglich.

#### Ernährungserhebung mittels Verzehrshäufigkeitsfragebogen

Ergänzend zu der prospektiven Verzehrserhebung mittels Wiegeprotokollen wird ein Verzehrshäufigkeitsfragebogen (FFQ) eingesetzt. Dieser erhebt den Lebensmittelverzehr retrospektiv über die vergangenen zwölf Monate. Der FFQ wurde eigens für eine pflanzenbasierte Ernährung am BfR in Zusammenarbeit mit der Universität Bonn entwickelt. Grundlage waren die Lebensmittellisten aus der RBVD-Studie des BfR [20], aus einer Doktorarbeit des Instituts für Ernährungsepidemiologie der Universität Bonn [67] sowie aus weiteren in früheren Studien eingesetzten FFQs [68, 69]. Der FFQ beinhaltet Lebensmittel, die im Rahmen einer veganen oder vegetarischen Ernährungsweise gehäuft verzehrt werden, wie pflanzliche Brotaufstriche, pflanzliche Milch-, Fleisch- und Fischalternativprodukte. Um zeitlichen Veränderungen in der Lebensmittelauswahl bei Mischköstlern ebenfalls gerecht zu werden, sind entsprechende Anpassungen erfolgt. Der FFQ fragt die Häufigkeit und Portionsgröße des Verzehrs von mehr als 150 Lebensmittel-Items ab. Die Studienteilnehmenden füllen den FFQ beim zweiten Besuch im Studienzentrum, am Standort Berlin zusätzlich am dritten Besuchstag, am PC aus.

Die Ergebnisse einer ersten Validierungsstudie zeigen, dass der für COPLANT entwickelte FFQ den Verzehr pflanzlicher Alternativprodukte mit einer guten Reliabilität und einer akzeptablen relativen Validität erhebt\*. Eine umfassende Validierung des FFQ, die alle Lebensmittelitems berücksichtigt, ist im Rahmen der Hauptstudie am BfR geplant.

<sup>\*</sup> Masterarbeit von Kira Tessel: Untersuchung der Reliabilität und Validität der Ernährungserhebung von pflanzlichen Alternativprodukten anhand eines neu entwickelten Verzehrshäufigkeitsfragebogens, BfR, 2023

Neben der Ernährung werden in der Basiserhebung der COPLANT-Studie eine Vielzahl an gesundheitsbezogenen Merkmalen erhoben, die als Auswirkungen pflanzenbasierter Ernährungsweisen (Endpunkte), als potentielle Confounder oder Mediatoren der Assoziationen pflanzenbasierter Ernährungsformen mit gesundheitlichen Endpunkten oder als Modifikatoren dieser Zusammenhänge von Interesse sind (Kapitel 6.3 bis 6.12).

#### 6.3 Anthropometrie

Die Körpergröße wird mit Stadiometern (Firma seca) gemessen. Taillen- und Hüftumfang werden mit einem Maßband (Firma seca) gemessen. Bei allen Messungen sind die Teilnehmenden barfuß und bis auf die Unterwäsche entkleidet. Das Körpergewicht wird im Rahmen der bioelektrischen Impedanzanalyse bestimmt.

#### 6.4 Bioelektrische Impedanzanalyse

Die bioelektrische Impedanzanalyse (BIA) ist eine Methode zur Bestimmung der Körperzusammensetzung. Die BIA basiert auf der Messung des elektrischen Widerstandes, den ein Körper einem elektrischen Wechselstrom entgegensetzt. Unter Berücksichtigung von Alter, Geschlecht, Körpergröße, Körpergewicht und Taillenumfang werden die fettfreie Masse und der Körperfettanteil berechnet. Es wird das Gerät mBCA 515 der Firma seca eingesetzt. Die Teilnehmenden stehen in Unterwäsche und barfuß in aufrechter Position auf dem Messgerät. Die Messung wird nicht durchgeführt bei schwangeren Frauen sowie Teilnehmenden mit Metallimplantaten, aktiven Prothesen oder Herzschrittmachern. Risiken bestehen für die Teilnehmenden nicht.

#### 6.5 Messung der Knochengesundheit

Die Knochengesundheit wird mittels quantitativem Ultraschall (QUS) am Fersenbein mit dem Gerät Inus S (Firma medical ECONET GmbH) bestimmt. An beiden Fersen werden jeweils zwei Messungen vorgenommen. Eine Messung dauert etwa zwei Minuten. Risiken bestehen für die Teilnehmenden nicht.

In einer Vorstudie am BfR mit acht Teilnehmenden und Einschluss aller für die Studie vorgesehenen Geräte wurde eine akzeptable Reliabilität der Messung verschiedener Knochenparameter nachgewiesen. Externe Studien zeigen, dass eine QUS-Messung an der Ferse mit in prospektiven Studien validierten Geräten eine Frakturrisikoabschätzung erlaubt [70].

#### 6.6 Blutdruckmessung

Der Blutdruck wird mit dem Gerät Boso carat professional (Firma BOSCH + SOHN GmbH u. Co. KG) im Sitzen gemessen. Der systolische und der diastolische Blutdruck sowie der Puls

werden jeweils dreimal im Abstand von zwei Minuten bestimmt. Vor der ersten Messung sollen die Teilnehmenden mindestens fünf Minuten ruhig gesessen haben.

#### 6.7 Akzelerometrie

Die Teilnehmenden tragen über einen Zeitraum von bis zu sieben Tagen den Aktivitätssensor Move 4 (Firma movisens GmbH). Dieser zeichnet die körperliche Aktivität kontinuierlich auf. Das Gerät wird den Teilnehmenden beim ersten Besuch im Studienzentrum ausgehändigt und bis zum zweiten Besuch zurückgegeben.

#### 6.8 Messung der Handgreifkraft

Die Handgreifkraft wird mittels des Dynamometers Jamar Plus+ Digital Hand Dynamometer (Firma Performance Health) an beiden Händen jeweils dreimal gemessen.

Die Handgreifkraft ist ein sehr guter Indikator für die allgemeine Muskelkraft. Aktuelle Erkenntnisse deuten darauf hin, dass die Messung der Handgreifkraft eine einfache Methode zur Beurteilung verschiedener Erkrankungs- und Sterberisiken darstellt [71].

#### 6.9 Weitere Untersuchungen

Jedes Studienzentrum kann weitere Untersuchungen in Abhängigkeit von lokalen Forschungsinteressen und Gerätekapazitäten durchführen. Diese Untersuchungen werden in den Ethikanträgen der einzelnen Studienzentren spezifiziert.

## 6.10 Erhebung der Einnahme von Arzneimitteln und Nahrungsergänzungsmitteln

Die Einnahme von Arzneimitteln und Nahrungsergänzungsmitteln in den letzten vier Wochen vor dem zweiten Besuchstermin wird in einem standardisierten Interview mit einem Instruments zur datenbankgestützten Online-Erfassung von Medikamentendaten (IDOM) [72] erhoben.

#### 6.11 Befragungen

Den Teilnehmenden werden Fragen zur Soziodemographie, zum Lebensstil, zur Ernährung, zu nachhaltigem Verhalten, zu Vorerkrankungen und sonstigen gesundheitlichen Merkmalen gestellt (Tabelle 2). Dafür wird ein computergestützter Selbstausfüllfragebogen eingesetzt.

**Tabelle 2** Übersicht über die Module des Fragebogens

| Modul | Inhalt |
|------------------|--------------------------|
| Soziodemographie | Alter |
| | Geschlecht |
| | Familienstand |
| | Haushaltsgröße und -form |

| Modul | Inhalt |
|---|---|
| | Anzahl Kinder |
| | Bildung |
| | Beruf |
| | Haushaltseinkommen |
| Lebensstil | Rauchstatus |
| | Alkoholkonsum |
| | Körperliche Aktivität |
| | Musikalische Aktivität |
| | Verwendung von Kosmetikprodukten |
| | Schlafqualität |
| | Chronotopie (nur in Berlin) |
| Ernährung | Ernährungsweise (Art, Dauer, Motivation) |
| | Mahlzeitenverhalten |
| | Verwendung von Jodsalz und Fluorid |
| Gesundheitsfragen | Diagnostizierte Krankheiten |
| | Diagnostizierte Allergien und Nahrungsmittelunverträglichkeiten |
| | Mentale Gesundheit |
| | Familienanamnese |
| | Fragen zur Frauengesundheit |
| | Fragen zu Mikrobiota |
| Nachhaltigkeit | Einkaufsverhalten und Außer-Haus-Verzehr |
| _ | Ausgaben für Lebensmittel |
| | Selbstversorgungsgrad |
| | Relevanz nachhaltiger Produkteigenschaften |
| | Soziale, kulturelle und gesellschaftliche Aspekte der Ernährung |
| | Einstellungen und Lebensführung |

#### 6.12 Sammlung von biologischen Proben

#### **Blutprobe**

Allen Studienteilnehmenden werden beim zweiten Untersuchungstermin nüchtern mindestens 54 ml Blut abgenommen. Die Blutentnahme sollte zwischen 7 und 10 Uhr erfolgen, um einen Einfluss der Tageszeit auf biologische Marker weitestgehend auszuschließen.

Einige Parameter (darunter Blutbild, Elektrolyte, Blutfette, Blutzucker, Leber- und Nierenwerte) werden unmittelbar in einem lokalen akkreditierten Labor bestimmt (Set 1, Anhang A2). Das übrige Blut (Set 2) wird fraktioniert und zum Teil bis zum Abschluss der Basiserhebung bei bis zu -80°C tiefgefroren, um mögliche Batcheffekte zu vermeiden. Am Universitätsklinikum Jena sollen ausgewählte Biomarker (Set 2A) zentral bestimmt und dort bis zum Ende der Basiserhebung auch Material für weitere Analysen (Set 2B) gelagert werden (Anhang A3). Optional kann an den einzelnen Standorten zusätzliches Blut für eine lokale Lagerung und spätere Analysen abgenommen werden (Set 3).

#### Urinprobe

Die Studienteilnehmenden sammeln am Vortag des zweiten Besuchstermins über 24 Stunden ihren Urin und bringen diesen am Besuchstag mit. Beim ersten Besuch erhalten die Teilnehmenden für die Sammlung des Urins Behälter und eine Anleitung (mündlich und schriftlich). Im Studienzentrum werden der gesamte 24-Stunden-Sammelurin gewogen und homogenisiert, der pH-Wert und optional das spezifische Gewicht bestimmt. Diese Informationen und der Sammelzeitpunkt werden protokolliert.

Einige Urinparameter werden unmittelbar in einem akkreditierten Labor bestimmt (Set 1). Der übrige Urin wird fraktioniert und bis zu den biochemischen Analysen nach Abschluss der Basiserhebung bei -80°C tiefgefroren. Ein Teil dieser Proben wird am Universitätsklinikum Jena für spätere Analysen gelagert (Set 2B, Anhang 3). Bei fehlendem Sammelurin wird im Studienzentrum eine Spontanurinprobe erbeten und für die Analysen des Set 1 und Set 2B genutzt. Optional können Fraktionen des Sammelurins und des Spontanurins am jeweiligen Studienzentrum lokal gelagert werden (Set 3).

#### Stuhlprobe

Die Studienteilnehmenden geben beim zweiten Besuch im Studienzentrum eine vollständige Stuhlprobe, die sie am Morgen zu Hause entnommen haben, ab. Alternativ kann die Stuhlprobe innerhalb von sieben Tagen nachgereicht werden. Für die Probennahme erhalten die Teilnehmenden beim ersten Besuch einen Sammelbehälter (Fecotainer) und eine Anleitung (mündlich und schriftlich). Die Stuhlproben werden am Untersuchungstag im Studienzentrum gewogen, eine Menge von 100 g homogenisiert und für die spätere Analyse aliquotiert. Die Zeitpunkte der Stuhlentnahme, der Ankunft im Studienzentrum, des Verarbeitungsbeginns und des Einfrierens sowie das Gewicht, die Beschaffenheit und der pH-Wert der Stuhlprobe werden protokolliert. Es werden 8 Aliquots je 1 g gesammelt. Diese sind vorgesehen für die Messung der Mikrobiota (Sequenzierung), SCFA, Gallensäuren, Calprotectin sowie 4 Rückstellproben. Die Stuhlproben werden kurzfristig im jeweiligen Studienzentrum und längerfristig am MRI bei -80°C bis zu den Analysen gelagert.

#### 7. Nachbeobachtung

#### Aktive Nachbeobachtung

Nach der Basiserhebung werden die Studienteilnehmenden alle drei bis fünf Jahre schriftlich kontaktiert und gebeten, Fragebögen auszufüllen (Abbildung 3). Damit sollen Veränderungen der Ernährungsweise, des Lebensstils und des Gesundheitszustandes erfasst werden. Im Rahmen dieser aktiven Nachbeobachtung wird auch das Neuauftreten ausgewählter Erkran-

kungen (darunter Typ 2 Diabetes, Herz-Kreislauf-Erkrankungen, Krebserkrankungen, Osteoporose) erhoben. Zur Verifizierung der Selbstangaben in den Fragebögen ist Einsichtnahme in Unterlagen der behandelnden Ärztin bzw. des behandelnden Arztes vorgesehen.

Bei erfolgreicher Einwerbung von Drittmitteln werden alle Studienteilnehmenden nach fünf bis zehn Jahren erneut ins Studienzentrum eingeladen. Teilnehmende, die nicht mehr in ihrer ursprünglichen Studienregion wohnen, werden ebenfalls eingeladen. Ihnen wird angeboten, das nächstgelegene Studienzentrum zu besuchen. Das Programm der Folgeuntersuchung wird im Wesentlichen dem der Basisuntersuchung entsprechen, um Veränderungen in interessierenden Merkmalen erfassen zu können.

#### Passive Nachbeobachtung

In COPLANT sollen Studiendaten mit Sekundärdaten zur gesundheitlichen Situation und Versorgung verknüpft werden. Bei auftretenden Erkrankungen wird ein Abgleich mit den Daten vorhandener epidemiologischer Register für Stoffwechselerkrankungen (z. B. Diabetes mellitus Typ 2), Herzinfarkt, Schlaganfall und Krebs angestrebt. Durch die Verknüpfung mit Abrechnungsdaten der gesetzlichen Krankenversicherung wird zudem die Grundlage für versorgungsepidemiologische und pharmakoepidemiologische Forschungsaktivitäten gelegt.

#### 8. Statistische Datenanalyse

#### 8.1 Statistische Methoden

Das multizentrische Design der Studie, in der Assoziationen von vier Ernährungsformen mit dem Auftreten von Krankheiten und Gesundheitsparametern untersucht werden, ist richtungsweisend für die geplanten statistischen Auswertungen. Wann immer möglich, werden die Auswertungen auf den Daten der gesamten Kohorte basieren. Wenn eine Fragestellung nur für eine bestimmte Teilpopulation von Interesse ist, werden entsprechende Teilkohorten gebildet. Das breite Spektrum an wissenschaftlichen Fragestellungen, das Studiendesign und die umfangreiche Datenerhebung erfordern die Anwendung von Methoden aus den Bereichen deskriptive und schließende Statistik [73], statistisch-epidemiologische Methoden [74], Machine Learning [75] und kausale Inferenz [76]. Für jedes Teilgebiet wird geeignetes statistisches und methodisches Fachwissen eingebracht, z. B. bioinformatische Methoden für die Verarbeitung und Analyse von Biomaterialien (Tabelle 3).

**Tabelle 3** Einsatz von statistischen Methoden in COPLANT

| Analysen | Beispiele |
|---|---|
| Querschnittsanalysen<br>(Daten der Basiserhebung) | <ul> <li>Deskriptive Statistik</li> <li>Zusammenhangsanalysen (Regressions- und Korrelationsanalysen)</li> <li>Prädiktive Modellierung mit Methoden des Machine Learnings</li> <li>Mustererkennungsverfahren (multivariate Verfahren, Machine Learning)</li> <li>Kausale Inferenz unter Modellierung kausaler Strukturen mit directed acyclic graphs (DAGs, DAG-based Regression)</li> </ul> |
| Analysen wiederholter Messungen (longitudinale Daten) | Gemischte lineare und nichtlineare Mo-<br>delle (mixed models) |
| Ereigniszeitanalysen (Analyse der Zeit bis zum Auftreten eines Ereignisses, z. B. einer Krankheit) | <ul> <li>Cox-Regression</li> <li>Parametrische Verfahren der Ereigniszeitanalyse</li> <li>Multistate-Modelle</li> <li>Competing Risk-Analyse</li> <li>Prädiktive Modellierung mit Methoden des Machine Learnings</li> <li>Kausale Überlebenszeitanalyse mit inverse probability weighting</li> </ul> |

Das multizentrische Design der Studie kann über geeignete Adjustierung oder Mehrebenenanalysen (multilevel modeling) bei der Datenanalyse berücksichtigt werden. Es kann angenommen werden, dass sich Beobachtungen (Studienteilnehmende) innerhalb eines Studienzentrums ähnlicher sind im Vergleich zu Beobachtungen außerhalb dieses Studienzentrums.
Im Rahmen von Mehrebenenanalysen kann diese Abhängigkeit der Beobachtungen modelliert
werden. Diese Modelle erlauben die Adjustierung für weitere Variablen, um beispielsweise
Confounding oder Effektmodifikation (Interaktion) zu adressieren.

Es ist davon auszugehen, dass sich Veganer, Vegetarier und Pescetarier neben der Ernährung in einer Vielzahl weiterer gesundheitsrelevanter Verhaltensweisen von Mischköstlern unterscheiden. Daraus resultiert eine komplexe Confoundersituation, die bei der Datenauswertung zu berücksichtigen ist.

#### 8.2 Planung des Stichprobenumfanges

Die Ermittlung des notwendigen Stichprobenumfanges basiert auf der Schätzung von 10-Jahres-Erkrankungsrisiken für den Vergleich der vier Ernährungsweisen. Dafür wurden publizierte Daten zu jährlichen Inzidenzen und relativen Risiken herangezogen. Als gesundheitliche Auswirkungen der pflanzenbasierten Ernährungsweisen wurden das Auftreten von Typ-2-Diabetes, Herz-Kreislauf-Erkrankungen und Krebs betrachtet. Es handelt sich dabei um häufige Volkskrankheiten, zu deren Vermeidung die Ernährung beitragen kann. Die Berechnungen erfolgten für die Gesamtkohorte mit acht geplanten Standorten.

#### 10-Jahres-Erkrankungsrisiken

Die jährliche Inzidenz von Typ-2-Diabetes, Herz-Kreislauf-Erkrankungen und Krebs lag zwischen 4 pro 1000 Personenjahre (0,4 %) für jüngere Altersgruppen (20 bis 50 Jahre) und 18 pro 1000 Personenjahre (1,8 %) für ältere Altersgruppen (etwa 50 Jahre und älter) [77-79]. Für den Vergleich von Vegetariern mit Mischköstlern wurden relative Erkrankungsrisiken von 0,63 (95% Konfidenzintervall: 0,54–0,74) für Diabetes [6], 0,75 (0,60–0,82) für ischämische Herzerkrankungen, 0,93 (0,86–1,00) für Herz-Kreislauf-Erkrankungen und 0,92 (0,87–0,98) für Krebs [5] berichtet.

Bei einer niedrigen jährlichen Inzidenz von 0,4 % sollten 1207 Personen pro Ernährungsform und damit insgesamt 4828 Personen in die Studie eingeschlossen werden, um ein relatives Risiko von 0,60 jeweils für den Vergleich der pflanzlichen Ernährungsweisen mit der gemischten Ernährungsform signifikant schätzen zu können (Alpha=0,05, Power=0,80, zweiseitiger Test).

Basierend auf diesen etwa 5000 Personen und 20 % Ausfällen bei der Nachbeobachtung wird eine Stichprobengröße von 6000 angestrebt. Daraus resultiert eine geplante Rekrutierung von im Mittel 750 (6000/8) Teilnehmenden pro Studienzentrum. Bei einer Ausfallquote von 28 % müssten 6400 Studienteilnehmende rekrutiert werden. Folglich würden jeweils zwischen 1500 und 1600 Studienteilnehmende in die vier Ernährungsgruppen eingeschlossen, wenn die Gesamtstichprobengröße zwischen 6000 und 6400 liegt.

#### Querschnittsanalysen zur Basiserhebung

Die geschätzte Stichprobengröße, die sich auf den Längsschnitt der Studie bezieht, ermöglicht im Querschnitt (Basiserhebung) genaue statistische Beschreibungen mit kleinen Konfidenzintervallen und entsprechende Gruppenvergleiche. Beispielsweise würde sich für einen mittleren Body-Mass-Index (BMI, kg/m²) von 25 kg/m² mit einer Standardabweichung von 5 kg/m² für eine der Ernährungsweisen (n=1600) ein enges 95%-Konfidenzintervall von 24,51 bis 25,49 (25 kg/m²  $\pm$  0,49 kg/m²) ergeben (Beispiel aus der RBVD-Studie: BMI für Veganer 22,9 kg/m²  $\pm$  3,2 kg/m² [20]). Ein geschätztes 95%-Konfidenzintervall für eine tägliche Gesamtenergieaufnahme (kcal/d) von 2000 kcal bei einer Standardabweichung von 150 kcal würde die Werte von 1985 bis 2015 kcal/d (2000 kcal/d  $\pm$  14,7 kcal/d) umfassen (Beispiel: Energieaufnahme 2270 kcal/d, 95%-Konfidenzintervall von 1800 bis 2762 kcal/d [20]).

Es ergibt sich zudem eine hohe statistische Power für Gruppenvergleiche, wenn der Stichprobenumfang für jede Ernährungsweise 1600 beträgt. Mit einem ungepaarten 2-Stichproben-t-Test kann beispielsweise ein Mittelwertsunterschied zwischen den Gruppen geprüft werden. Für den BMI kann ein mittlerer Unterschied von 0,6 kg/m² (angenommene Standardabweichung für den mittleren Unterschied von 4 kg/m²) bzw. für die Gesamtenergieaufnahme ein

mittlerer Unterschied von 70 kcal (angenommene Standardabweichung für den mittleren Unterschied von 500 kcal) statistisch signifikant nachgewiesen werden (Alpha=0,05, statistische Power = 80%, zweiseitiger Test).

#### 9. Nachhaltigkeitsanalyse

Um die Auswirkungen der betrachteten Ernährungsweisen in den Dimensionen Gesundheit, Umwelt, Gesellschaft und Wirtschaft zu untersuchen, wird eine Nachhaltigkeitsanalyse durchgeführt (in konzeptioneller Anlehnung an [80, 81]). Ziel ist es, ökologische, soziale und ökonomische Folgen der Ernährungsweisen zu analysieren und diese mit den Erkenntnissen zu gesundheitlichen Wirkungen zusammenzuführen. Die Basis für die Analysen in den einzelnen Dimensionen bilden die Erhebungen des Lebensmittelverzehrs mit der NutriDiary-App und dem FFQ (Kapitel 6.2), die Fragebogenmodule zu Ernährung, Verhalten im Alltag und Soziodemographie (Tabelle 3) sowie vertiefende Interviews mit mindestens acht Studienteilnehmenden (zwei Interviews pro Ernährungsweise) pro Studienzentrum. Ein Interview dauert etwa 90 Minuten und kann im Studienzentrum oder über Webkonferenz stattfinden.

Ökologische Auswirkungen werden über Lebenszyklusanalysen (Ökobilanz) ermittelt. Die betrachteten Wirkungskategorien umfassen insbesondere klimaschädliche Emissionen (ausgedrückt in CO<sub>2</sub>-Äquivalenten) und Primärenergieeinsatz, aber auch weitere indikative Angaben wie Wasserverbrauch, Landnutzung und den Product Environmental Footprint (PEF)-Indikator. Der PEF oder Umweltfußabdruck von Lebensmitteln ist ein auf mehreren Kriterien basierendes Maß für die Umweltleistung eines Produktes entlang seines Lebenswegs und aggregiert 13 Wirkungsindikatoren (z. B. CO<sub>2</sub>-Fußabdruck, Wasser- und Landnutzung, Versauerung) in einem Single-Score nach einer auf EU-Ebene vereinbarten Methode [82-84]. Den Ausgangspunkt der Analysen bilden der Lebensmittelverzehr der entsprechenden Ernährungsweise und dessen Auswirkungen von der Primärproduktion über die Verarbeitung bis zum Handel. Soweit möglich, werden Aspekte des Ernährungsverhaltens wie Einkaufsverhalten, Zubereitungsart, Lagerung und Nachbereitung (z. B. Entstehung von Lebensmittelabfällen) bei der Untersuchung ökologischer Auswirkungen berücksichtigt. Sachbilanzdaten (Life Cycle Inventory) werden z. B. den Ökobilanzdatenbanken Ecoinvent [85] und Agribalyse [86] entnommen.

Bei der Untersuchung **sozialer Auswirkungen** werden zum einen soziale Aspekte des Ernährungsverhaltens untersucht. Dazu gehören z. B. der Verzehr fair und tierwohlverträglich hergestellter Lebensmittel, die Esssituation sowie mit Ernährung in Verbindung stehende soziale Teilhabe bzw. Ausgrenzung, kulturelle Vielfalt und gesellschaftliches Engagement. Zum anderen werden Motivationen und Wertehaltungen (z. B. Bedeutung ethischer Aspekte) sowie allgemeiner Lebensstil der Teilnehmenden erforscht.

Die ökonomischen Auswirkungen werden primär über die mit den verschiedenen Ernährungsweisen direkt verbundenen Kosten auf Haushaltsebene betrachtet. Dabei werden insbesondere die Ausgaben für Lebensmittel berücksichtigt. Weitere Faktoren wie sozioökonomische Merkmale, Selbstversorgungsgrad, Preissensibilität und Relevanz von Verkaufsaktionen werden, soweit möglich, in die Analysen integriert. Indirekte Kosten der Ernährungsweisen werden in Form externer Umweltkosten bei Produktion und Verarbeitung zumindest abgeschätzt. Die Umweltkosten werden simultan zur Ökobilanzierung betrachtet.

Die Auswertungsmethoden im Feld der integrativen Nachhaltigkeitsbetrachtung werden stetig weiterentwickelt. Ein wichtiges Ziel der Nachhaltigkeitsanalyse ist es, neben der inhaltlichen Forschung ein Bewertungsinstrument mit Blick auf Ernährungsweisen zu entwickeln und anzuwenden. Aufgrund der Kombination von Methoden und Datenquellen wird ein breites Spektrum an Ergebnissen, von quantitativen (insbesondere Abschätzung ökologischer und ökonomischer Auswirkungen) bis hin zu semiquantitativen und qualitativen Aussagen (insbesondere Abschätzung sozialer Auswirkungen) generiert werden.

#### 10. Modul "Schwangere und Stillende"

## 10.1 Wissenschaftliche Fragestellungen des Moduls "Schwangere und Stillende"

Im Modul "Schwangere und Stillende" sollen in einem explorativen Ansatz mögliche Auswirkungen der Ernährungsweise der Mutter auf den Verlauf der Schwangerschaft und Stillzeit sowie die Entwicklung des Kindes innerhalb der ersten zwei Lebensjahre untersucht werden. Folgende wissenschaftliche Fragestellungen stehen im Vordergrund:

- 1. Ändern sich die Ernährungsweise und die Supplementierung von Nährstoffen während der Schwangerschaft und Stillzeit?
- 2. Wie sind Schwangere und Mütter mit unterschiedlicher Ernährungsweise hinsichtlich Soziodemographie, Lebensstil, Anthropometrie, Gesundheitszustand und Schwangerschaftsmerkmalen charakterisiert?
- 3. Hängen Stillinitierung, Stilldauer, Stillintensität sowie Zeitpunkt der Einführung und Art der Beikost von der Ernährungsweise der Mutter ab?
- 4. Ändert sich die Ernährungsweise der Mutter ein bzw. zwei Jahre nach der Geburt im Vergleich zur Stillzeit?
- 5. Ernähren sich vegan, vegetarisch bzw. pescetarisch ernährende Mütter ihre Kinder ebenfalls vegan, vegetarisch bzw. pescetarisch?

#### 10.2 Teilnehmerinnen am Modul "Schwangere und Stillende"

Das Modul "Schwangere und Stillende" soll an den Standorten Berlin, Karlsruhe, Jena und Gießen durchgeführt werden. Es sollen insgesamt etwa 800 Teilnehmerinnen im gebärfähigen

Alter (jeweils 100 Frauen in den Altersgruppen 18 bis 29 Jahre und 30 bis 39 Jahre pro Studienzentrum) rekrutiert werden. Bei etwa 772.000 Geburten [87] auf 10 Millionen Frauen im gebärfähigen Alter in Deutschland im Jahr 2021 [88] könnte bei 800 Teilnehmerinnen rein rechnerisch von ca. 60 Schwangeren zum Zeitpunkt der Rekrutierung ausgegangen werden. Tatsächlich könnte diese Zahl jedoch aufgrund des erwarteten höheren sozioökonomischen Status der Studienteilnehmerinnen im Vergleich mit der deutschen Allgemeinbevölkerung geringer ausfallen. Zudem ist nicht vorhersehbar, wie häufig sich Schwangere tatsächlich für eine Studienteilnahme interessieren. Dies könnte entscheidend von zielgruppenspezifischer Werbung für die Studie abhängen.

#### 10.3 Untersuchungsproramm des Moduls "Schwangere und Stillende"

Schwangere und Stillende können jeweils einmal an einem reduzierten Untersuchungsprogramm teilnehmen. Die Teilnehmerinnen werden zu vier Zeitpunkten untersucht:

- Zeitpunkt 1: 30. bis 35. Schwangerschaftswoche (3. Trimenon der Schwangerschaft)
- Zeitpunkt 2: drei bis vier Monate nach der Geburt (postpartum)
- Zeitpunkt 3: ein Jahr nach der Geburt
- Zeitpunkt 4: zwei Jahre nach der Geburt.

Zu den Zeitpunkten 1, 2 und 4 wird in das Studienzentrum eingeladen. Zu Zeitpunkt 3 wird zu Hause ein Fragebogen ausgefüllt.

Frauen, die zum Zeitpunkt der Rekrutierung schwanger sind und an der COPLANT-Studie teilnehmen möchten, werden in der 30. bis 35. Schwangerschaftswoche erstmals in das Studienzentrum eingeladen. Die Teilnehmerinnen protokollieren wie die übliche COPLANT Teilnehmenden an vier Tagen ihre Ernährung mittels der NutriDiary-App und füllen einen webbasierten FFQ aus (Kapitel 6.2). Sie sammeln einen 24-Stunden-Urin und entnehmen eine Stuhlprobe (Kapitel 6.12). Im Studienzentrum werden Nüchternblut entnommen, das Körpergewicht und der Blutdruck der Schwangeren bestimmt. Unter Verwendung des im Hauptprogramm eingesetzten Fragebogens (Tabelle 3) ergänzt um Fragen aus anderen Studien an Schwangeren (z.B. PEACHES) wird ein für die Schwangerschaft spezifischer Fragebogen entwickelt und eingesetzt. Zusätzlich werden Daten aus dem Mutterpass (darunter Gewicht zu Beginn der Schwangerschaft und Gewichtszunahme im Verlauf) erhoben.

Drei bis vier Monate nach der Geburt des Kindes werden die Frauen zu einem zweiten Besuch eingeladen. Frauen, die zum Zeitpunkt der Rekrutierung bereits geboren haben und stillen, werden drei bis vier Monate nach der Geburt erstmals untersucht. Es wird ein für die Lebensphase spezifischer Fragebogen (unter anderem mit Fragen zu Geburt, Beginn und Dauer des Stillens) eingesetzt. Weitere Informationen zur Geburt (darunter Gestationsalter und Geburtsmodus) werden dem Mutterpass, Informationen zur Entwicklung des Kindes (darunter Geburtsgewicht und -größe, postnatale Gewichts- und Größenentwicklung, Auffälligkeiten in der

Entwicklung) dem Kinderuntersuchungsheft entnommen. Zusätzlich zu den bereits genannten Bioproben wird um eine Muttermilchprobe gebeten.

Ein Jahr nach der Geburt des Kindes erhalten die Frauen einen webbasierten Fragebogen, der unter anderem Fragen zu Stilldauer und Beikost enthält. Zwei Jahre nach der Geburt werden unter anderem Daten zur Gewichts- und Größenentwicklung sowie Auffälligkeiten in der Entwicklung des Kindes erhoben. Frauen, die nach diesem Kurzprogramm weiter an CO-PLANT teilnehmen möchten, können zwei Jahre nach der Geburt das Hauptprogramm der Studie durchlaufen.

Frauen, die nach der Teilnahme am Hauptprogramm der Basiserhebung schwanger werden, werden gebeten, dies ihrem Studienzentrum mitzuteilen, so dass sie zusätzlich in das Modul "Schwangere und Stillende" aufgenommen werden können.

#### 11. Modul "Kids & Family"

#### 11.1 Wissenschaftliche Fragestellungen des Moduls "Kids & Family"

Im Modul "Kids & Family" werden an den Standorten Berlin und Karlsruhe zusätzlich die Kinder der erwachsenen Studienteilnehmenden untersucht. Die daraus resultierende dyadische Datenstruktur (Mutter/Vater-Kind-Paare) wird genutzt, um Einflüsse des familiären Ernährungsumfeldes auf das Ernährungsverhalten der Kinder zu erforschen.

Das Modul "Kids & Family" kann wegen der geringen Stichprobengröße (Kapitel 11.2) und fehlender Bioproben nicht alle relevanten Forschungsfragen in absehbarer Zeit umfassend adressieren. Es fokussiert daher auf eine Auswahl an Fragestellungen im familiären Ernährungskontext, die zunächst im Querschnitt explorativ untersucht werden, um darauf aufbauend Hypothesen zu generieren. Neben dem inhaltlichen Wissen sollen auch methodische Erkenntnisse gewonnen werden, anhand derer eine Ausweitung des Moduls auf andere COPLANT-Studienzentren geprüft werden kann. Bei ausreichender Teilnehmendenzahl und vorhandener Finanzierung wird eine Nachbeobachtung angestrebt.

Das Modul "Kids & Family" adressiert zunächst folgende Forschungsthemen:

- Untersuchung der Kinder von Eltern mit pflanzenbasierter bzw. omnivorer Ernährungsweise hinsichtlich:
  - o Ernährungsweise: Art (vegan, vegetarisch, pescetarisch oder omnivor) und Dauer
  - Lebensmittelverzehr und N\u00e4hrstoffsupplementierung
  - o Größe, Gewicht und Körperzusammensetzung
- Untersuchung von Verhaltensdeterminanten, die potenzielle Zusammenhänge zwischen den Ernährungsweisen von Kindern und Eltern erklären könnten:
  - soziale Verhaltensdeterminanten (darunter Ernährungsweisen innerhalb der Familie,
     Familienmahlzeiten und Lebensmittelangebot, soziale Normen)

- psychologische Verhaltensdeterminanten (darunter Autonomie und Wahlmöglichkeiten der Kinder, Modellverhalten)
- Untersuchung von Aspekten des Studiendesigns einschließlich der Rekrutierung, insbesondere:
  - Anteil an erwachsenen COPLANT-Studienteilnehmenden mit minderjährigen Kindern
  - Altersstruktur der potenziell zu rekrutierenden Kinder (einschließlich derjenigen ohne Studieneinwilligung)
  - Teilnahmebereitschaft der Kinder der erwachsenen Studienteilnehmenden, insgesamt und in Abhängigkeit von der Ernährungsweise

Die aus Public-Heath-Perspektive hoch relevante Untersuchung der Auswirkungen einer im Kindesalter beginnenden vegetarischen oder veganen Ernährungsweise unter anderem auf Nährstoffstatus, Wachstum, kognitive Entwicklung und Knochenmineralisierung ist aufgrund des Designs des Moduls "Kids & Family" derzeit nicht möglich. Diese Fragen müssen auf der Basis vorhandener longitudinaler Datenerhebungen adressiert werden, um zeitnah Erkenntnisse hierzu zu gewinnen. Deshalb werden weiterführende Analysen im Rahmen der Mutter-Kind-Kohorte Programming of Enhanced Adiposity Risk in CHildhood - Early Screening (PEACHES) vorgeschlagen [89].

#### 11.2 Teilnehmende am Modul "Kids & Family"

Die erwachsenen COPLANT-Teilnehmenden werden über das Modul "Kids & Family" informiert und gefragt, ob sie mit einem oder mehreren im selben Haushalt lebenden Kind bzw. Kindern daran teilnehmen möchten. In Deutschland leben in etwa 20 % der Haushalte minderjährige Kinder [90, 91]. Durch die Adressierung von Familien bei der Rekrutierung wird erwartet, dass dieser Anteil unter den erwachsenen COPLANT-Teilnehmenden bei 30 bis 40 % liegt. Bei jeweils etwa 800 teilnehmenden Erwachsenen an den Standorten Berlin und Karlsruhe wird bei einem Anteil an Kindern von etwa 35 % und einer erwarteten Beteiligung von 50 bis 75 % (EsKiMo II-Studie: 59 % [92]; KiESEL-Studie: 75 bis 82 % [59]) pro Standort mit 140 bis 210 teilnehmenden Kindern im Alter von 0 bis 17 Jahren gerechnet. Damit werden an jedem Standort etwa 35 bis 50 Kinder je Ernährungsgruppe des teilnehmenden Elternteils erwartet.

#### 11.3 Untersuchungsprogramm des Moduls "Kids & Family"

Erwachsende COPLANT-Studienteilnehmende mit minderjährigen Kindern werden in Berlin und Karlsruhe eingeladen, zusätzlich am Modul "Kids & Family" teilzunehmen. Mit den Eltern wird ein gemeinsamer Termin im Studienzentrum vereinbart.

In einem Basisfragebogen geben die Eltern Auskunft zur familiären Situation einschließlich der Essgewohnheiten und relevanten sozialen und psychologischen Verhaltensdeterminanten (Abbildung 7). Der Fragebogen beinhaltet außerdem Fragen zu Soziodemografie, Lebensstil und Gesundheit der Kinder. Weitere Daten werden in Abhängigkeit vom Alter der Kinder erhoben: Bei Kindern unter 11 Jahren beantwortet der teilnehmende Elternteil weitere Fragen. Diese beinhalten unter anderem den Lebensmittelverzehr der Kinder, der mit einem FFQ der Studie zur Gesundheit von Kindern und Jugendlichen in Deutschland (KiGGS) [93] und zusätzlichen Fragen zu pflanzlichen Alternativprodukten erhoben wird. Kinder ab 11 Jahren beantworten die weiteren Fragen selbst. Dieses Vorgehen und der Grenzwert für die Bildung der Altersgruppen orientieren sich an Datenerhebungen bei Kindern und Jugendlichen in KiGGS [94]. Für Kinder unter 3 Jahren beantworten die Eltern Fragebögen, die unter anderem für das Modul "Schwangere und Stillende" entwickelt wurden und Daten zum Stillen, zur Beikost und zum Übergang zur Familienkost erheben. Bei allen Kindern werden Körpergröße und Körpergewicht gemessen. Bei Kindern ab 5 Jahren werden zusätzlich die Körperzusammensetzung mittels BIA (Berlin und Karlsruhe) sowie der Blutdruck und die Knochengesundheit mittels Ultraschall am Fersenbein (nur Berlin) bestimmt.

Im Anschluss an diese Basiserhebung werden die Eltern gefragt, ob sie zu einer Nachbeobachtung (Berlin und Karlsruhe) und zu weiterführenden Untersuchungen, wie dem Führen von Ernährungsprotokollen und qualitativen Methoden (nur Berlin), bereit wären.



**Abbildung 7** Design des COPLANT-Moduls "Kids & Family"

BIA = Bioelektrische Impedanzanalyse, FFQ = Food Frequency Questionnaire, KiGGS = Studie zur Gesundheit von Kindern und Jugendlichen in Deutschland. †Am Standort Berlin werden bei Kindern

ab 5 Jahren zusätzlich Blutdruckmessungen und eine Untersuchung der Knochengesundheit mittels Ultraschall durchgeführt.

#### 12. Qualitätsmanagement

Das Design der COPLANT-Studie stellt eine Herausforderung an die Vergleichbarkeit der generierten Daten sowohl zwischen den beteiligten Studienzentren als auch zwischen den geplanten Erhebungswellen (Basiserhebung, Nachbeobachtungen) dar. Zur Gewährleistung einer höchstmöglichen Datenqualität, die dem Anspruch der Vergleichbarkeit zwischen Studienzentren und Erhebungswellen genügt, wird ein Qualitätsmanagementkonzept erarbeitet. Das Konzept orientiert sich an den Anforderungen der Guten Wissenschaftlichen und Epidemiologischen Praxis [95] sowie an Qualitätsstandards für epidemiologische Kohortenstudien [96] unter Abwägung von Nutzen und Aufwand.

Kernpunkte des Qualitätsmanagements der COPLANT-Studie sind:

- (1) eine standardisierte Datenerhebung in allen Studienzentren, die durch die Verwendung einheitlicher Erhebungsinstrumente und Arbeitsanweisungen (SOPs) sowie regelmäßige Schulungen und Zertifizierungen des Studienpersonals gewährleistet wird
- (2) Kontrollen der Struktur-, Prozess- und Ergebnisqualität über regelmäßige Monitorings
  - a. der Studienzentren (auf Ausstattung und Organisation; Strukturqualität)
  - b. der Rekrutierung und Datenerhebung (auf SOP-Konformität; Prozessqualität)
  - c. der Daten und Dokumente (auf Rekrutierungserfolg innerhalb festgelegter Strata sowie auf Vollständigkeit und Plausibilität der erhobenen Daten; Ergebnisqualität)
- (3) fehlerminimierende Dateneingaben durch automatisierte Prüfungen auf fehlende Angaben und plausible Wertebereiche
- (4) halbjährliche bzw. jährliche Qualitätsberichte an das Konsortium und Abstimmung von Qualitätssicherungsmaßnahmen bei Handlungsbedarf (z. B. problematische Rekrutierung innerhalb einzelner Strata).

Detaillierte Anforderungen an das Qualitätsmanagement und Maßnahmen zu deren Umsetzung sind dem gesonderten Qualitätsmanagementkonzept zu entnehmen.

#### 13. Datenschutz, Informationssicherheit und Datenmanagement

In der COPLANT-Studie erfolgt die Erhebung und Verarbeitung von personenbezogenen Daten (alle Informationen, die sich auf eine identifizierte oder identifizierbare natürliche Person beziehen) zum Zweck des oben dargelegten Forschungsvorhabens in Übereinstimmung mit der DSGVO und auf Grundlage der Einwilligungen (DSGVO Art. 6 Abs. 1 lit. a und Art. 9 Abs. 1 lit. a). Alle im Rahmen der COPLANT-Studie erhobenen personenbezogenen Daten der Studienteilnehmenden werden streng vertraulich behandelt. Grundlage der Datenverarbeitung ist

eine zwischen den Studienzentren geschlossene Vereinbarung über gemeinsame Verantwortlichkeit gemäß Art. 26 Abs. 1 S. 1 DSGVO. Zudem sind jedes Studienzentrum und deren Mitarbeitende an die datenschutzrechtlichen Vereinbarungen ihres jeweiligen Institutes gebunden.

#### 13.1 Arten personenbezogener Daten

Im Rahmen der COPLANT-Studie werden die in Tabelle 4 gelisteten Arten von personenbezogenen Daten erhoben und verarbeitet.

**Tabelle 4** Arten personenbezogener Daten

| Art der Daten | Informationen und Zweck |
|---|---|
| Personenidentifizierende Daten | Name, Vornamen, Wohnanschrift(en), Telefonnummer(n) und E-Mail-Adresse(n) zum Zweck der Kontaktierung und Vereinbarung von Terminen |
| Weitere identifizierende Daten | Name und IK- bzw. Registernummer der Krankenversicherung,<br>Krankenversichertennummer zum Zweck der Erhebung von Se-<br>kundärdaten |
| | Altersbereich, Geschlecht, Ernährungsform zum Zweck der Zu-<br>ordnung von Teilnehmenden zu Rekrutierungsstrata |
| Verwaltungsdaten | Dokumentation von Terminvereinbarungen, Kontaktversuchen, Kontaktergebnissen zum Zweck der Teilnehmendenbetreuung sowie der Optimierung von Prozessen und der Beteiligung |
| Forschungsdaten | Pseudonymisierte Daten aus Befragungen, (körperlichen) Untersuchungen, Bioproben (Blut, Urin, Stuhl, Speichel) sowie Laborparameter zum Zweck der wissenschaftlichen Auswertung |
| Sekundär- und Registerdaten | externe, nicht im Rahmen der COPLANT-Studie erhobene Forschungsdaten (Gesundheits- und Sozialdaten) von Krankenkassen und aus Registern zum Zweck der Nachverfolgbarkeit von Erkrankungen u.a. |

#### 13.2 Übergeordnete Prinzipien

Umfang und Charakter der erhobenen Daten sowie ihre zentralisierte und automatisierte Verarbeitung stellen höchste Anforderungen an den Schutz dieser Daten. Jede beteiligte Institution stellt sicher, dass die Datenerhebung und der Umgang mit den Daten in Übereinstimmung mit der DSGVO erfolgen. Der Datenschutz und die Informationssicherheit werden während aller Phasen des Projekts konzeptionell sichergestellt und permanent überprüft. Bei der Erhebung, Speicherung und Verwaltung der personenidentifizierenden Daten und Forschungsdaten gelten als übergeordnete Prinzipien die Vertraulichkeit, die Trennung von personenidentifizierenden Daten und Forschungsdaten, die Pseudonymisierung der Forschungsdaten, die Verhinderung ungewollter Re-Identifizierung der Teilnehmenden sowie die Datensicherheit. Eine Re-Identifizierung von Teilnehmenden wird nur in bestimmten, klar definierten Fällen not-
wendig sein, beispielsweise um die Teilnehmenden mit mitteilungswürdigen Befunden zu kontaktieren. Dabei wird darauf geachtet, Daten nur in dem Umfang freizugeben, in dem sie zur Erreichung des jeweiligen Ziels unbedingt erforderlich sind. Durch organisatorische Maßnahmen wird sichergestellt, dass außerhalb der Studienzentren keine unautorisierten Personen Zugriff auf personenbezogene Daten der COPLANT-Studie erhalten.

#### 13.3 Organisationsstruktur aus Sicht des Datenmanagements

Die Anforderungen an den Datenschutz und die Informationssicherheit erfordern, dass personenidentifizierende Daten und Verwaltungsdaten getrennt von pseudonymisierten Forschungsdaten erhoben und verarbeitet werden. Entsprechend dieser Anforderung und aufgrund des multizentrischen Designs der COPLANT-Studie wurden die in Abbildung 8 visualisierte Organisationsstruktur und Datenflüsse etabliert.



Abbildung 8 Organisationsstruktur und Datenflüsse der COPLANT-Studie

An jedem der beteiligten Institute ist ein Studienzentrum angesiedelt. Ein Studienzentrum besteht aus dem Teilnahmemanagement und dem Untersuchungszentrum. Aus Gründen des Datenschutzes sollen das Teilnahmemanagement und das Untersuchungszentrum auf physischer, technischer und personeller Ebene getrennt sein. Unter dem Gesichtspunkt der Verhältnismäßigkeit kann in den einzelnen Studienzentren jedoch von einer personell-organisatorischen Trennung abgesehen werden. Bei der Kontaktierung und dem Empfang der Teilnehmenden in den Studienzentren sowie bei den Befragungen und Untersuchungen kann es da-

her zu personellen Überschneidungen kommen. Durch technische Maßnahmen (Nutzung unterschiedlicher PCs) und räumliche Trennung sollte jedoch eine getrennte Erhebung und Verarbeitung von Kontaktdaten und pseudonymisierten Forschungsdaten sichergestellt sein.

Die Erhebung von personenidentifizierenden Daten und Verwaltungsdaten erfolgt durch das Teilnahmemanagement der Studienzentren mittels der lokal implementierten Teilnahmemanagementsoftware webMODYS. Aus Gründen der Effizienz, Standardisierung und Kosteneinsparung wurden zudem am BfR eine zentrale Treuhandstelle (THS) und ein zentrales Datenmanagement eingerichtet. In der THS werden personenidentifizierende Daten getrennt von und ohne direkte Verknüpfung mit den pseudonymisierten Forschungsdaten langfristig in der THS-Datenbank gespeichert. Die THS-Datenbank basiert auf der Software E-PIX (https://www.ths-greifswald.de/forscher/e-pix/) und ist auf einem geschützten Server am BfR implementiert. Des Weiteren verwaltet die THS die Einwilligungs- und Datenschutzerklärungen der Teilnehmenden mittels der THS-Software gICS (https://www.ths-greifswald.de/forscher/gics/), welche ebenfalls auf einem geschützten Server des BfR implementiert ist. Die Übertragung von personenidentifizierenden Daten sowie Einwilligungs- und Datenschutzerklärungen und deren Speicherung in der THS erfolgen durch das jeweilige Teilnahmemanagement mittels gesicherter Internetverbindungen (VPN-Tunnel, Zertifikatsdateien, Benutzerlogin). Der Zugriff zur THS ist auf namentlich benanntes und autorisiertes Personal beschränkt. Die Erhebung, Speicherung und Verwaltung der pseudonymisierten Forschungsdaten erfolgt mittels REDCap (https://www.project-redcap.org/) in der COPLANT-Forschungsdatenbank. REDCap ist eine Web-Applikation zur Erstellung und Verwaltung von Online-Umfragen und Datenerfassungsbögen, insbesondere für epidemiologische und klinische Forschungsprojekte. Die COPLANT-Forschungsdatenbank und die REDCap-Web-Applikation sind auf einem geschützten Server des BfR implementiert, getrennt von der THS-Datenbank. Die Forschungsdatenbank wird durch das Datenmanagement am BfR verwaltet. Die Erhebung und Speicherung der pseudonymisierten Forschungsdaten erfolgt über gesicherte Internetverbindungen (VPN-Tunnel, Zertifikatsdateien, Benutzerlogin) per Webbrowser und ist auf namentlich benanntes, autorisiertes Personal beschränkt.

Rohdaten, die nicht unmittelbar in der Forschungsdatenbank gespeichert werden können, werden auf einer Nextcloud-Dateiablage (<a href="https://nextcloud.com/de/">https://nextcloud.com/de/</a>) des BfR abgelegt. Die Dateiablage ist auf geschützten Server des BfR implementiert. Der Zugriff zur Dateiablage durch die Untersuchungszentren erfolgt über gesicherte Internetverbindungen (VPN-Tunnel, Zertifikatsdateien, Benutzerlogin) per Webbrowser und ist auf namentlich benanntes, autorisiertes Personal beschränkt.

#### 13.4 Pseudonymisierung

Zur Wahrung des Rechts auf informationelle Selbstbestimmung ist zu gewährleisten, dass aus der Verarbeitung der erhobenen Daten keine Rückschlüsse auf individuelle Verhältnisse einer einzelnen natürlichen Person gezogen werden können. Dafür ist es notwendig, den Umfang der erhobenen und verarbeiteten Daten auf das zur Durchführung der Studie erforderliche Minimum zu beschränken, personenidentifizierende Daten und Forschungsdaten stets getrennt voneinander zu speichern und zu verarbeiten sowie alle Forschungsdaten zu pseudonymisieren. Zu diesem Zweck wird jedem Teilnehmenden eine Teilnahmenummer (TN-ID) und eine Studiennummer (Study-ID) zugewiesen. Die TN-ID wird als Identifier im Teilnahmemanagement und in der THS verwendet. Die Study-ID ist mit der TN-ID in einer Liste verknüpft. Die Study-ID wird im Untersuchungszentrum verwendet, um die Forschungsdaten pseudonymisiert zu speichern. Im Falle von Widerrufen oder mitteilungswürdigen Befunden können die pseudonymisierten Forschungsdaten mittels der Verknüpfung von Study-ID und TN-ID den jeweiligen Teilnehmenden zugeordnet werden. Die Liste mit der Verknüpfung der TN-ID und Study-ID ist nur berechtigten Personen des Teilnahmemanagements, der THS und den Leitern der Studienzentren zugänglich. Das Teilnahmemanagement und die zentrale THS haben keinen direkten Zugriff auf die pseudonymisierten Forschungsdaten.

#### 13.5 Aufbewahrungsfristen

Personenbezogene Daten müssen gelöscht werden, wenn sie nicht mehr gebraucht werden, um die spezifische Funktion zu erfüllen. Zur Erfüllung des Zwecks der COPLANT-Studie ist 20 eine langfristige Datenspeicherung voraussichtlich bis 30 Jahren von (Nachbeobachtungszeit) erforderlich. Die personenidentifizierenden Daten werden nach dem Ende der Nachbeobachtungszeit der Studie gelöscht (gemäß DSGVO) oder wenn kein weiterer direkter Kontakt zu den Teilnehmenden und keine Re-Identifizierung von Teilnehmenden mehr erforderlich sind. Daraus ergibt sich eine Speicherdauer für die personenidentifizierenden Daten von mindestens 20 bis 30 Jahren. In diesem Zeitraum ist eine regelmäßige Aktualisierung der personenidentifizierenden Daten vorgesehen (Vitalstatus, Kontaktadresse, Telefonnummer, Familienname etc.).

Die in der Studie erhobenen Forschungsdaten werden langfristig und pseudonymisiert in der Forschungsdatenbank gespeichert. Die Dauer der Speicherung ergibt sich aus dem Zweck der Studie und dem daraus unmittelbar folgenden Zeitraum der wissenschaftlichen Auswertung der Forschungsdaten.

Daten, die die COPLANT-Studie von externen Quellen (z. B. von Krankenversicherungen) erhält und Forschungsdaten, die die COPLANT-Studie für wissenschaftliche Auswertungen zur Verfügung gestellt hat, können nicht vor Ablauf der Aufbewahrungsfristen, die sich aus der

Guten Epidemiologischen Praxis ergeben, gelöscht werden. Im Fall eines entsprechenden Widerrufs werden die Zuordnungslisten der Pseudonyme gelöscht und die archivierten Übergabedaten des widerrufenden Teilnehmenden damit anonymisiert.

Papierdokumente (Barcodes, Laufzettel etc.), die für den Besuch im Studienzentrum notwendig sind, werden im Studienzentrum unter Einhaltung der erforderlichen Sicherheitsmaßnahmen zum Schutz vor Verlust und unbefugter Einsichtnahme in abschließbaren Aktenschränken verwahrt. Unmittelbar nach dem Besuch und der Datenübermittlung werden nicht länger benötigte Papierdokumente datenschutzgerecht vernichtet.

#### 13.6 Datennutzung, Datenweitergabe und Datenempfänger

Die Nutzung der erhobenen Forschungsdaten und Bioproben innerhalb des COPLANT-Konsortiums ist in der Nutzungsordnung geregelt. Die Projektverwaltung des zentralen Datenmanagements koordiniert die Nutzungsanträge bzw. -anzeigen. Der wissenschaftliche Lenkungsausschuss, bestehend aus den Leiterinnen und Leitern der Studienzentren, prüft die Anträge und entscheidet über die Nutzung der Daten.

Es erfolgt nur eine Datenweitergabe von pseudonymisierten Forschungsdaten. Datenempfänger sind Partner der COPLANT-Studie und assoziierte Partner. Zudem haben Teilnehmende die Möglichkeit, einer potenziellen Datenweitergabe an Forschungspartner, die aus Ländern innerhalb der EU, Ländern mit Angemessenheitsbeschluss außerhalb der EU und an Forschungspartner in Drittländern außerhalb der EU ohne Angemessenheitsbeschluss zuzustimmen. Für die Datenweitergabe muss jeweils eine Einwilligungserklärung der Teilnehmenden vorliegen und mit den Forschungspartnern muss, soweit für das Land kein Angemessenheitsbeschluss vorliegt, ein Vertrag zur Absicherung des Drittlandtransfers abgeschlossen werden. Aktuell ist kein Drittlandtransfer geplant.

## 14. Ethik

#### 14.1 Ethische Grundsätze

Die COPLANT-Studie wird in Übereinstimmung mit dem Grundgesetz, dem Bundesdatenschutzgesetz, den einschlägigen Landesdatenschutzgesetzen, den Meldegesetzen der Bundesländer, dem Krebsregistergesetz und der Deklaration von Helsinki des Weltärztebundes durchgeführt. Dabei gelten folgende Grundsätze:

- Vorrang der Rechte und des Wohlergehens der Teilnehmenden vor allen anderen Interessen einschließlich der Forschungsziele
- freiwillige Teilnahme nach Aufklärung

- Respektierung kultureller Unterschiede im gesamten Verlauf der Studie, von der Rekrutierung über die Gewinnung der Daten und Bioproben bis zu ihrer wissenschaftlichen Nutzung
- Beachtung des besonderen Schutzes von vulnerablen Studienteilnehmenden
- Transparenz der Vorgehensweise, Finanzierung, institutioneller Verbindungen und möglicher Interessenskonflikte
- datenschutzgerechtes Erheben, Verarbeiten und Nutzen personenbezogener Daten
- Einhaltung technischer und organisatorischer Maßnahmen zur Sicherstellung der Vertraulichkeit, Verfügbarkeit und Integrität der gespeicherten Informationen (Informationssicherheit)
- Einhaltung der Prinzipien der Guten Epidemiologischen Praxis [95] im gesamten Forschungsprozess.

## 14.2 Aufklärung und Einwilligung

Die Teilnahme an der COPLANT-Studie ist freiwillig. Die informierte Einwilligung in die Studienteilnahme wird in Form der Einwilligungserklärung dokumentiert. Die Ablehnung der Teilnahme führt für die eingeladenen Personen nicht zu Nachteilen.

Nachdem sie die Studieninformation zu Hause gelesen haben, werden die Studieninteressenten im Studienzentrum von Ärztinnen und Ärzten der COPLANT-Studie oder angemessen qualifizierten Mitarbeitenden aufgeklärt. Die aufklärende Person muss sich davon überzeugen, dass die Studieninteressentin bzw. der Studieninteressent verstanden hat, wozu er seine Einwilligung gibt. Das für die Aufklärung und Einholung der Einwilligungserklärung zuständige Personal ist darin geschult und handelt nach den detaillierten Anweisungen einer SOP.

Da es unmöglich ist, alle zukünftigen Forschungsfragen im Detail vorherzusehen, wird die Einwilligungserklärung so gestaltet, dass ein möglichst breites Forschungsfeld offengehalten wird. Dies beinhaltet auch die Analyse von biologischen und genetischen Markern in Blutproben und weiteren Bioproben gemäß den Zielen der COPLANT-Studie.

Die Teilnehmenden werden unter anderem darüber aufgeklärt,

- dass die Teilnahme an der COPLANT-Studie freiwillig und kostenlos ist.
- dass die Laufzeit der COPLANT-Studie auf mindestens 20 Jahre angelegt ist.
- wie lange ihre Einwilligungen gültig sein werden.
- dass die Einwilligungen auch bei Verlust der Selbstbestimmungsfähigkeit und nach dem Tod des Teilnehmenden gültig bleiben.
- dass die Teilnahme keine Untersuchung durch eine Ärztin oder einen Arzt ersetzt und die mitgeteilten Ergebnisse keine medizinischen Befunde oder ärztlichen Diagnosen sind.

- dass personenidentifizierende Daten streng getrennt von den Forschungsdaten in den Studienzentren gehalten und ausschließlich für die Kontaktaufnahme verwendet werden. Forschungsdaten werden ausschließlich pseudonymisiert gespeichert und ausgewertet.
- dass die Daten und Bioproben langfristig gespeichert bzw. gelagert und für zukünftige Forschungsfragen zu Ernährung und häufigen Volkskrankheiten genutzt werden. In Zukunft können Szenarien auftreten, die den Einsatz neuer Methoden oder die Ausweitung der ursprünglichen Forschungsfragen bedingen, z. B. aufgrund neuer Techniken oder Erkenntnisse, die zu Beginn der Studie noch nicht definiert oder unbekannt waren. Die Einwilligung der Teilnehmenden umfasst auch die Nutzung ihrer Daten und Bioproben für diese Zwecke. Die Ziele der COPLANT-Studie bleiben dabei unverändert.
- dass die Nutzung der Daten und Bioproben entsprechend der Nutzungsordnung der Studie erfolgt. Diese regelt die Weitergabe von Daten und Bioproben an Forscher im In- und Ausland.
- dass die Teilnehmenden das Recht haben, jederzeit über die über sie gespeicherten Daten Auskunft zu verlangen.
- dass die Teilnehmenden das Recht haben, ihre Einwilligungserklärung jederzeit ohne Angabe von Gründen schriftlich zu widerrufen.

Die Teilnehmenden werden nach der Aufklärung gebeten, einzuwilligen,

- dass sie sich dazu bereiterklären, am Untersuchungs- und Befragungsprogramm der COPLANT-Studie teilzunehmen.
- dass sie mit der langfristigen Speicherung, Verarbeitung, Nutzung und Überlassung ihrer Daten an andere Forscher einverstanden sind.
- dass sie sich dazu bereiterklären, Bioproben abzugeben bzw. abnehmen zu lassen.
   Die Bioproben können nur abgegeben und gewonnen werden, wenn die Teilnehmenden die Eigentumsrechte an den Bioproben vorbehaltlich ihres allgemeinen Persönlichkeitsrechts an das jeweilige Studienzentrum übertragen.
- dass weitere Gesundheitsdaten, einschließlich Krankheitsdiagnosen und Behandlungsinformationen, von ihrer Hausärztin bzw. ihrem Hausarzt oder anderen behandelnden Ärztinnen bzw. Ärzten angefordert werden dürfen. Das ist notwendig, da die Teilnehmenden diese Informationen häufig selbst nicht präzise wissen oder fachgerecht widergeben können. Dafür werden die Teilnehmenden um die Angabe von Namen und Praxisadresse ihrer Hausärztin bzw. ihres Hausarztes oder weiterer behandelnder Ärztinnen und Ärzte im ambulanten Bereich sowie in Krankenhäusern gebeten.

Die Teilnehmenden werden gebeten, die behandelnden Ärztinnen und Ärzte von der Schweigepflicht zu entbinden.

- dass ihr Vitalstatus regelmäßig überprüft wird und im Todesfall Angaben zu Ort, Zeit und Ursachen von den Meldebehörden, Gesundheitsämtern und behandelnden Ärztinnen und Ärzten angefragt werden dürfen.
- dass weitere Gesundheits- und Sozialdaten, die für wissenschaftliche Zwecke benötigt werden, von externen Datenquellen angefordert werden dürfen. Hierfür werden die Teilnehmenden gebeten, den Namen ihrer Krankenversicherung und ihre Krankenversichertennummer anzugeben. Diese Angaben werden nur zeitlich befristet und ausschließlich in der unabhängigen Treuhandstelle gespeichert. Gesundheits- und Sozialdaten hingegen werden pseudonymisiert übermittelt und den Forschungsdaten zugeordnet. Die Einzelheiten dieser Prozesse sind im Datenschutzkonzept beschrieben.
- dass sie in regelmäßigen Intervallen (per Brief, E-Mail, Telefon oder Internet) erneut kontaktiert und interviewt (und in diesem Kontext wieder identifiziert) werden, um Informationen über Änderungen in ihrem Lebensstil und anderen Risikofaktoren sowie über aufgetretene Erkrankungen zu erhalten.
- dass sie nach etwa fünf bis zehn Jahren zu mindestens einer Folgeuntersuchung eingeladen werden.

Für das Modul "Kids & Family" gelten besondere Befragungsrichtlinien für Minderjährige. Daher werden angepasste Studieninformationen und Einwilligungserklärungen in leicht zugänglicher Form sowie in klarer und einfacher Sprache erarbeitet und verwendet. Die Einwilligungserklärung muss bei jüngeren Kindern von beiden Erziehungsberechtigten, bei Kindern bzw. Jugendlichen ab 14 Jahren zusätzlich vom Kind selbst unterschrieben werden.

#### 14.3 Widerrufsrecht

Jeder Teilnehmende selbst bzw. seine gesetzliche Vertreterin oder sein gesetzlicher Vertreter hat jederzeit das Recht und die Möglichkeit, seine Einwilligungserklärung ohne Angabe von Gründen ganz oder teilweise zu widerrufen. Dem Teilnehmenden entstehen dadurch keine Nachteile. Der Widerruf muss in schriftlicher Form gegenüber dem für den Studienteilnehmenden zuständigen Teilnahmemanagement erfolgen. Falls der Teilnehmende bei der Erklärung seines Widerrufs Hilfe benötigt, kann er sich an das für ihn zuständige Teilnahmemanagement wenden und von dort z. B. ein einfaches Widerrufsformular erhalten. Unterschiedliche Reichweiten des Widerrufs sind möglich:

#### Kein weiterer Kontakt

Der oder die Teilnehmende wird nicht weiter kontaktiert. Personenidentifizierenden Daten, die nicht zur Umsetzung weiterer Widerrufsrechte (z. B. Widerruf der Nutzung von Forschungsdaten) benötigt werden, werden gelöscht. Die erhobenen Forschungsdaten und Bioproben bleiben jedoch erhalten und dürfen weiterhin für die Forschung genutzt werden. Ebenso dürfen Informationen aus sekundären Datenquellen eingeholt werden.

## Kein weiterer Zugang, aber weitere Nutzung

Der oder die Teilnehmende wird nicht weiter kontaktiert. Personenidentifizierenden Daten, die nicht zur Umsetzung weiterer Widerrufsrechte (z. B. Widerruf der Nutzung von Forschungsdaten) benötigt werden, werden gelöscht. Die erhobenen Forschungsdaten und Bioproben bleiben erhalten und dürfen weiterhin für die Forschung genutzt werden. Es werden jedoch keine weiteren Informationen aus sekundären Datenquellen eingeholt.

#### Keine weitere Nutzung

Der oder die Teilnehmende wird nicht weiter kontaktiert. Die personenidentifizierenden Daten werden gelöscht. Es werden keine weiteren Daten eingeholt. Bereits gesammelte Forschungsdaten und Bioproben werden gesperrt und stehen für zukünftige Forschungsfragen nicht zu Verfügung. Daten aus bereits durchgeführten Analysen können nicht nachträglich gelöscht werden. Auf Verlangen des Teilnehmenden können jedoch seine Bioproben vernichtet werden.

#### 14.4 Risiken bei Befragungen und Untersuchungen

Das Risikopotenzial der Befragungen und Untersuchungen ist insgesamt gering. Möglicherweise werden einzelne Fragen im Fragebogen oder im Interview als unangenehm empfunden. Die Teilnehmenden können jedoch Fragen, die sie nicht beantworten können oder möchten, mit "weiß nicht" oder "keine Angabe" beantworten. Alle medizinischen Untersuchungen und Entnahmen von Bioproben werden von geschultem, zertifiziertem und erfahrenem Personal durchgeführt. Nach der Blutabnahme besteht ein geringes Risiko, dass an der Einstichstelle ein Bluterguss (Hämatom), eine leichte Entzündung oder eine Infektion entsteht. In sehr seltenen Fällen kann es passieren, dass ein Nerv verletzt wird. Die Probanden werden darüber aufgeklärt, dass bei Untersuchungen auch bisher unentdeckte Erkrankungen und Auffälligkeiten gefunden werden können, die eine weitere Abklärung bedürfen und ggf. als Belastung empfunden werden können. Die Studienteilnehmenden können selbst entscheiden, ob sie diese erfahren möchten. Bei am Modul "Kids & Family" teilnehmenden minderjährigen Kindern werden nur nicht-invasive Erhebungsmethoden verwendet und keine Bioproben gesammelt.

#### 14.5 Möglicher Nutzen für die Teilnehmenden

Die Teilnehmenden an COPLANT helfen vor allem, wertvolle Daten für die bevölkerungsbezogene Forschung zu pflanzlich basierten Ernährungsweisen bereitzustellen. Die erhobenen Daten können jedoch auch der bzw. dem Teilnehmenden selbst zugutekommen.

Wichtige Ergebnisse der Untersuchungen werden den Teilnehmenden bereits im Studienzentrum mitgeteilt. Die Ergebnisse der Labormessungen werden ihnen in einem Brief zugesandt.
Bei Laborbefunden außerhalb der Referenzwerte werden die Teilnehmenden von der Studienärztin bzw. dem Studienarzt telefonisch kontaktiert. Falls es sinnvoll ist, aufgrund der Ergebnisse eine Ärztin bzw. einen Arzt aufzusuchen, werden die Teilnehmenden darauf hingewiesen. Das genaue Vorgehen bei der Ergebnismitteilung regelt eine SOP.

Die Studienteilnahme ist dennoch nicht mit einem Gesundheits-Check gleichzusetzen. Es werden keine medizinischen Befunde erhoben und keine ärztlichen Diagnosen gestellt.

#### 14.6 Versicherung für die Teilnehmenden und Aufwandsentschädigung

Eine generelle (verschuldensunabhängige) Teilnahmeversicherung ist aufgrund des geringen Risikopotenzials der Studie und wegen des möglichen Nutzens einer Teilnahme nicht vorgesehen. Für schuldhaft verursachte Schäden haften die Verantwortlichen des Studienzentrums. Im Schadensfall übernimmt deren Haftpflichtversicherung diese Haftung. Für die Teilnahme wird eine Wege-Unfallversicherung abgeschlossen.

Die Teilnehmenden erhalten eine monetäre Aufwandsentschädigung, eine Küchenwaage sowie Befunde aus der Untersuchung im Studienzentrum sowie dem Basislabor. Dies zielt darauf ab, die Idee des Spendens von Daten und Bioproben für die Forschung zu Prävention und Behandlung von Volkskrankheiten zu stärken. Daten und Bioproben sollen als allgemeines Gut angesehen werden.

#### 15. Wissenschaftlicher Beirat

Zur Begleitung der COPLANT-Studie wird ein wissenschaftlicher Beirat mit Expertinnen und Experten aus verschiedenen wissenschaftlichen Disziplinen eingesetzt. Es ist vorgesehen, dass der wissenschaftliche Beirat den Lenkungsausschuss der COPLANT-Studie auf Sitzungen zweimal im Jahr berät. Folgende Expertinnen und Experten haben ihre Bereitschaft zur Mitarbeit im wissenschaftlichen Beirat erklärt und werden dazu eingeladen:

- Prof. Dr. Phillipp Wild, Klinische Epidemiologie, Universitätsmedizin Mainz (Epidemiologie und Prävention von kardiovaskulären Erkrankungen)
- Prof. Dr. Matthias Schulze, Molekulare Epidemiologie, Deutsches Institut für Ernährungsforschung, Bergholz-Rehbrücke (Ernährungsepidemiologie, Epidemiologie und Prävention von Typ 2 Diabetes)

- Prof. Dr. Kristin Junge, School für Health und Social Sciences, AKAD Hochschule Stuttgart (Humanernährung und Toxikologie)
- Prof. Dr. Alexander Moschen, Universität Linz (Gastroenterologie und Hepatologie, Mikrobiom)
- Prof. Dr. Juliana Raupp, Institut für Publizistik- und Kommunikationswissenschaft, Fachbereich Politik- und Sozialwissenschaften, Freie Universität Berlin (Organisationskommunikation, Politische Kommunikation)
- Prof. Dr. Nina Langen, Fachgebiet Bildung für Nachhaltige Ernährung und Lebensmittelwissenschaft, Technische Universität Berlin (Agrarökonomie, nachhaltiger Konsum, Lebensmittelverschwendung)
- Prof. Ulrich Mansmann, Institut für Biometrie und Epidemiologie, Ludwig-Maximilians-Universität München (Expertise im Bereich Kinderstudien und Daten)

#### Referenzen

- Allensbach I. Anzahl der Personen in Deutschland, die sich selbst als Vegetarier einordnen oder als Leute, die weitgehend auf Fleisch verzichten, von 2014 bis 2019. [cited 2020 28.07.2020]; Available from: <a href="https://de.statista.com/statistik/daten/studie/173636/umfrage/lebenseinstellung-anzahl-vegetarier/">https://de.statista.com/statistik/daten/studie/173636/umfrage/lebenseinstellung-anzahl-vegetarier/</a>.
- 2. Allensbach II. Personen in Deutschland, die sich selbst als Veganer einordnen oder als Leute, die weitgehend auf tierische Produkte verzichten, in den Jahren 2015 bis 2019. [cited 2020 28.07.2020]; Available from: <a href="https://de.statista.com/statistik/daten/studie/445155/umfrage/umfrage-in-deutschland-zur-anzahl-der-veganer/">https://de.statista.com/statistik/daten/studie/445155/umfrage/umfrage-in-deutschland-zur-anzahl-der-veganer/</a>.
- 3. BMEL. Forsa-Befragung des Bundeslandwirtschaftsministeriums zu Fleischkonsum / Ernährungsverhalten. 2020 11.06.2020]; Available from: <a href="https://www.bmel.de/SharedDocs/Meldungen/DE/Presse/2020/200524-">https://www.bmel.de/SharedDocs/Meldungen/DE/Presse/2020/200524-</a> fleischkonsumernaehrungsverhalten.html.
- 4. Le, L.T. and J. Sabate, *Beyond meatless, the health effects of vegan diets: findings from the Adventist cohorts.* Nutrients, 2014. **6**(6): p. 2131-47.
- 5. Dinu, M., et al., Vegetarian, vegan diets and multiple health outcomes: a systematic review with meta-analysis of observational studies. Crit Rev Food Sci Nutr, 2016: p. 0.
- 6. Papier, K., et al., Vegetarian diets and risk of hospitalisation or death with diabetes in British adults: results from the EPIC-Oxford study. Nutrition & Diabetes, 2019. **9**(1): p. 7.
- 7. Richter, M., et al., *Vegan diet. Position of the German Nutrition Society (DGE)*. Ernahrungs Umschau, 2016. **63**(05): p. M262.
- 8. Gehring, J., et al., Consumption of Ultra-Processed Foods by Pesco-Vegetarians, Vegetarians, and Vegans: Associations with Duration and Age at Diet Initiation. The Journal of Nutrition, 2020.
- 9. Blume, K., et al., Aufnahme von Umweltkontaminanten über Lebensmittel (Cadmium, Blei, Quecksilber, Dioxine und PCB). Ergebnisse des Forschungsprojektes LExUKon. 2010, Bundesinstitut für Risikobewertung.
- 10. Schwarz, M.A., et al., *Cadmium exposure from food: the German LExUKon project.* Food Additives & Contaminants: Part A, 2014. **31**(6): p. 1038-1051.
- 11. Schwarz, M.A., et al., *Dioxin and dl-PCB exposure from food: the German LExUKon project*. Food Addit Contam Part A Chem Anal Control Expo Risk Assess, 2014. **31**(4): p. 688-702.
- 12. Krajcovicová-Kudládková, M., et al., *Cadmium blood concentrations in relation to nutrition*. Cent Eur J Public Health, 2006. **14**(3): p. 126-9.
- 13. Tong, T.Y.N., et al., Risks of ischaemic heart disease and stroke in meat eaters, fish eaters, and vegetarians over 18 years of follow-up: results from the prospective EPIC-Oxford study. Bmj, 2019. **366**: p. 14897.
- 14. Iguacel, I., et al., *Veganism, vegetarianism, bone mineral density, and fracture risk: a systematic review and meta-analysis.* Nutr Rev, 2019. **77**(1): p. 1-18.
- 15. Iguacel, I., et al., *Vegetarianism and veganism compared with mental health and cognitive outcomes: a systematic review and meta-analysis.* Nutr Rev, 2020.
- 16. Appleby, P.N. and T.J. Key, *The long-term health of vegetarians and vegans.* Proc Nutr Soc, 2016. **75**(3): p. 287-93.
- 17. Leitzmann, C., R. Schönhöfer-Rempt, and M. Boy, *Ernährung und Gesundheit von Vegetariern.*Die Giessener Vegetarier-Studie. Echo-Verlag Hannover, 1988: p. 9-14.
- 18. Waldmann, A., et al., *Dietary intakes and lifestyle factors of a vegan population in Germany:* results from the German Vegan Study. Eur J Clin Nutr, 2003. **57**(8): p. 947-55.

- 19. Dawczynski, C., et al., Nutrient Intake and Nutrition Status in Vegetarians and Vegans in Comparison to Omnivores the Nutritional Evaluation (NuEva) Study. Front Nutr, 2022. 9: p. 819106.
- 20. Weikert, C., et al., *Vitamin and Mineral Status in a Vegan Diet.* Dtsch Arztebl Int, 2020. **117**(35-36): p. 575-582.
- 21. Rubner-Institut, M. Nationales Ernährungsmonitoring Durchführung und Auswertung von repräsentativen Erhebungen zu Lebensmittelverzehr, Energie- und Nährstoffzufuhr, Ernährungsstatus und weiteren Aspekten des Ernährungsverhaltens der Bevölkerung in Deutschland. 24.10.2023]; Available from: <a href="https://www.mri.bund.de/de/institute/ernaehrungsverhalten/forschungsbereiche/nationales-ernaehrungsmonitoring/">https://www.mri.bund.de/de/institute/ernaehrungsverhalten/forschungsbereiche/nationales-ernaehrungsmonitoring/</a>.
- 22. Avnon, T., et al., *The impact of a vegan diet on pregnancy outcomes.* J Perinatol, 2021. **41**(5): p. 1129-1133.
- 23. Kesary, Y., K. Avital, and L. Hiersch, *Maternal plant-based diet during gestation and pregnancy outcomes*. Arch Gynecol Obstet, 2020. **302**(4): p. 887-898.
- 24. Wang, Z., et al., Effects of Dietary Patterns during Pregnancy on Preterm Birth: A Birth Cohort Study in Shanghai. Nutrients, 2021. **13**(7): p. 2367.
- 25. Piccoli, G.B., et al., *Vegan–vegetarian diets in pregnancy: danger or panacea? A systematic narrative review.* BJOG: An International Journal of Obstetrics & Gynaecology, 2015. **122**(5): p. 623-633.
- 26. Forsa, Ernährungsreport 2022 Ergebnisse einer repräsentativen Bevölkerungsbefragung. 2022.
- 27. Patelakis, E., et al., *Prevalence of vegetarian diet among children and adolescents in Germany. Results from EsKiMo II.* Ernaehrungs Umschau, 2019. **66**(5): p. 85-91.
- 28. Grant, R., et al., *Cardiovascular disease risk factors profile among australian vegetarian and nonvegetarian teenagers.* Am J Lifestyle Med, 2021. **15**(3): p. 313-321.
- 29. Hovinen, T., et al., *Vegan diet in young children remodels metabolism and challenges the statuses of essential nutrients.* EMBO Molecular Medicine, 2021. **13**(2): p. e13492.
- 30. Desmond, M.A., et al., *Growth, body composition, and cardiovascular and nutritional risk of 5-to 10-y-old children consuming vegetarian, vegan, or omnivore diets.* The American Journal of Clinical Nutrition, 2021. **113**(6): p. 1565-1577.
- 31. Mokhtari, E., et al., Association between plant-based diets and metabolic health status in adolescents with overweight and obesity. Scientific Reports, 2022. **12**(1): p. 13772.
- 32. Ambroszkiewicz, J., et al., *Bone status and adipokine levels in children on vegetarian and omnivorous diets*. Clinical Nutrition, 2019. **38**(2): p. 730-737.
- 33. Elliott, L.J., et al., *Vegetarian diet, growth, and nutrition in early childhood: A longitudinal cohort study.* Pediatrics, 2022. **149**(6).
- 34. Jensen, C.F., Vitamin B12 levels in children and adolescents on plant-based diets: A systematic review and meta-analysis. Nutrition Reviews, 2022.
- 35. Weder, S., et al., Energy, macronutrient intake, and anthropometrics of vegetarian, vegan, and omnivorous children (1–3 Years) in Germany (VeChi Diet Study). Nutrients, 2019. **11**(4): p. 832.
- 36. Michaelson, V., K.A. Pilato, and C.M. Davison, *Family as a health promotion setting: A scoping review of conceptual models of the health-promoting family.* PLOS ONE, 2021. **16**(4): p. e0249707.
- 37. Dallacker, M., R. Hertwig, and J. Mata, *The frequency of family meals and nutritional health in children: A meta-analysis.* Obesity Reviews, 2018. **19**(5): p. 638-653.
- 38. Dallacker, M., R. Hertwig, and J. Mata, *Quality matters: A meta-analysis on components of healthy family meals.* Health Psychology, 2019. **38**(12): p. 1137-1149.
- 39. Knobl, V., et al., *Happy and healthy: How family mealtime routines relate to child nutritional health.* Appetite, 2022. **171**: p. 105939.
- 40. Frank, M., et al., *Prevalence and temporal trends of shared family meals in Germany. Results from EsKiMo II.* Ernahrungs Umschau, 2019. **66**(4): p. 60-67.

- 41. Peters, A., et al., Framework and baseline examination of the German National Cohort (NAKO). Eur J Epidemiol, 2022. **37**(10): p. 1107-1124.
- 42. Allès, B., et al., Comparison of Sociodemographic and Nutritional Characteristics between Self-Reported Vegetarians, Vegans, and Meat-Eaters from the NutriNet-Santé Study. Nutrients, 2017. **9**(9): p. 1023.
- 43. Bradbury, K.E., T.Y.N. Tong, and T.J. Key, *Dietary Intake of High-Protein Foods and Other Major Foods in Meat-Eaters, Poultry-Eaters, Fish-Eaters, Vegetarians, and Vegans in UK Biobank.* Nutrients, 2017. **9**(12).
- 44. Willett, W., et al., Food in the Anthropocene: the EAT-Lancet Commission on healthy diets from sustainable food systems. Lancet, 2019. **393**(10170): p. 447-492.
- 45. Grosso, G., et al., *Nutrition in the context of the Sustainable Development Goals*. European journal of public health, 2020. **30**(Suppl\_1): p. i19-i23.
- 46. Union, E., Farm to Fork Strategy For a fair, healthy and environmentally-friendly food system. 2020: Brussel.
- 47. (WBGU), W.B.d.B.G.U., Welt im Wandel Gesellschaftsvertrag für eine Große Transformation. Wissenschaftlicher Beirat der Bundesregierung Globale Umweltveränderungen 2011: Berlin.
- 48. FAO, et al., The State of Food Security and Nutrition in the World 2020. Transforming food systems for affordable healthy diets. 2020, FAO: Rome.
- 49. HLPE, Food security and nutrition: building a global narrative towards 2030. A report by the High Level Panel of Experts on Food Security and Nutrition of the Committee on World Food Security. 2020: Rome.
- 50. Wissenschaftlicher Beirat für Agrarpolitik, E.u.g.-c.V.b.B.W., *Politik für eine nachhaltigere Ernäh-rung: Eine integrierte Ernährungspolitik entwickeln und faire Ernährungsumge-bungen gestalten*. 2020: Berlin.
- 51. Godfray, H.C.J., et al., *Meat consumption, health, and the environment.* Science, 2018. **361**(6399).
- 52. Jetzke, T.R., S.; Keppner, B.; Domröse, L.; Wunder, S.; Ferrari, A., *Die Zukunft im Blick: Fleisch der Zukunft. Trendbericht zur Abschätzung der Umweltwirkungen von pflanzlichen Fleischersatzprodukten, essbaren Insekten und In-vitro-Fleisch.* 2019, Umweltbundesamt (UBA): Dessau-Roßlau.
- 53. Mbow, C., et al., Food Security, in Climate Change and Land: an IPCC special report on climate change, desertification, land degradation, sustainable land management, food security, and greenhouse gas fluxes in terrestrial ecosystems. 2019, Intergovernmental Panel on Climate Change.
- 54. Nelson, M.E., et al., *Alignment of Healthy Dietary Patterns and Environmental Sustainability: A Systematic Review.* Adv Nutr, 2016. **7**(6): p. 1005-1025.
- 55. Springmann, M., et al., *Analysis and valuation of the health and climate change cobenefits of dietary change.* Proc Natl Acad Sci U S A, 2016. **113**(15): p. 4146-51.
- 56. Reineke, A., Pigeot, I., Ahrens, W., Rach, S., MODYS—A Modular Control and Documentation System for Epidemiological Studies. Instruments for Health Surveys in Children and Adolescents, Springer Series on Epidemiology and Public Health, ed. K. Bammann, Lissner, L., Pigeot, I., Ahrens, W. (eds) 2019: Springer
- 57. Enzenbach, C., et al., Evaluating selection bias in a population-based cohort study with low baseline participation: the LIFE-Adult-Study. BMC Med Res Methodol, 2019. **19**(1): p. 135.
- 58. Kroke, A., et al., *The DONALD Study. History, current status and future perspectives.* Eur J Nutr, 2004. **43**(1): p. 45-54.
- 59. Nowak, N., et al., *KiESEL The Children's Nutrition Survey to Record Food Consumption for the youngest in Germany.* BMC Nutrition, 2022. **8**(1): p. 64.
- 60. Wark, P.A., et al., Validity of an online 24-h recall tool (myfood24) for dietary assessment in population studies: comparison with biomarkers and standard interviews. BMC Med, 2018. **16**(1): p. 136.

- 61. Eldridge, A.L., et al., Evaluation of New Technology-Based Tools for Dietary Intake Assessment-An ILSI Europe Dietary Intake and Exposure Task Force Evaluation. Nutrients, 2018. **11**(1).
- 62. Authority, E.F.S., General principles for the collection of national food consumption data in the view of a pan-European dietary survey. EFSA Journal 2009. **7**(12).
- 63. Authority, E.F.S., Guidance on the EU Menu methodology. 2014: EFSA Journal. p. 3944.
- 64. Carroll, R.J., et al., *Taking advantage of the strengths of 2 different dietary assessment instruments to improve intake estimates for nutritional epidemiology.* Am J Epidemiol, 2012. **175**(4): p. 340-7.
- 65. Freedman, L.S., et al., Combining a Food Frequency Questionnaire With 24-Hour Recalls to Increase the Precision of Estimation of Usual Dietary Intakes-Evidence From the Validation Studies Pooling Project. Am J Epidemiol, 2018. **187**(10): p. 2227-2232.
- 66. *NutriDiary: Innovative Ernährungserhebung für wissenschaftliche Studien*. 16.11.2023]; Available from: <a href="https://www.nutridiary-app.de/">https://www.nutridiary-app.de/</a>.
- 67. Freese, J.A., *A 24-hour food list for dietary assessment in large-scale epidemiological studies.* 2005, Rheinische Friedrich-Wilhelms-Universität Bonn.
- 68. Dyett, P., et al., Evaluation of a validated food frequency questionnaire for self-defined vegans in the United States. Nutrients, 2014. **6**(7): p. 2523-2539.
- 69. Max Rubner-Institut, Nationale Verzehrsstudie II. Ergebnisbericht Teil 2 2008: Karlsruhe.
- 70. V., D.O.e., Prophylaxe, Diagnostik und Therapie der Osteoporose bei postmenopausalen Frauen und bei Männern. Leitlinie des Dachverbandes der deutschsprachigen wissenschaftlichen osteologichen Gesellschaften e. V.. Langfassung

2017.

- 71. López-Bueno, R., et al., *Thresholds of handgrip strength for all-cause, cancer, and cardiovascular mortality: A systematic review with dose-response meta-analysis*. Ageing Res Rev, 2022. **82**: p. 101778.
- 72. Mühlberger N, B.C., Stark R, Holle R, *Datenbankgestützte Online-Erfassung von Arzneimitteln im Rahmen gesundheitswissenschaftlicher Studien Erfahrungen mit der IDOM-Software.* Informatik, Biometrie und Epidemiologie in Medizin und Biologie, 2003. **34**(4): p. 601-611.
- 73. J., H. and S. L., *Angewandte Statistik Methodensammlung mit R*. 2016, Heidelberg: Springer.
- 74. Rothman, K. and T. Lash, *Modern Epidemiology*. 4 ed. 2020: Lippincott Williams & Wilkins.
- 75. Gareth, J., et al., An Introduction to Statistical Learning. 2013: Springer New York.
- 76. Hernán, M. and J. Robins, Causal Inference: What If. 2020: Chapman & Hall/CRC.
- 77. Tamayo, T., et al., *The Prevalence and Incidence of Diabetes in Germany*. Dtsch Arztebl Int, 2016. **113**(11): p. 177-82.
- 78. (Hrsg), R.K.-I., Gesundheit in Deutschland. Gesundheitsberichterstattung des Bundes. Gemeinsam getragen von RKI und Destatis., RKI, Editor. 2015: Berlin.
- 79. Koch-Institut, R., Krebs in Deutschland für 2015/2016, in Robert Koch-Institut (Hrsg) und die Gesellschaft der epidemiologischen Krebsregister in Deutschland e.V. (Hrsg). 2019: Berlin.
- 80. Hoffmann, I., Verschiedene Ernährungsweisen: integrativ und mehrdimensional bewertet. , in Ernährungsökologie. Komplexen Herausforderungen integrativ begegnen., I.S. Hoffmann, K.; Leitzmann, C., Editor. 2011, oekom Verlag: München. p. 38-45.
- 81. Schneider, K.H., I.; Leitzmann, C. , *Ernährungsökologie Komplexen Herausforderungen integrativ begegnen*, in *Spiegel der Forschung*. 2012: Justus-Liebig Universität Gießen. p. 44-53.
- 82. European Commission, 2013/179/EU. Empfehlung der Kommission vom 9. April 2013 für die Anwendung gemeinsamer Methoden zur Messung und Offenlegung der Umweltleistung von Produkten und Organisationen. 2013: Brussels, Belgium.
- 83. European Commission, *Product Environmental Footprint Pilot Guidance. Guidance for the implementation of the EU Product Environmental Footprint (PEF) during the Environmental Footprint (EF) pilot phase: Version 5.2 February 2016.* 2016: Brussels, Belgium.

- 84. European Commission, *PEFCR Guidance document, Guidance for the development of Product Environmental Footprint Category Rules (PEFCRs), version 6.3, May 2018.* . 2018: Brussels, Belgium.
- 85. Ecoinvent, ecoinvent Database. <a href="https://ecoinvent.org/">https://ecoinvent.org/</a>.
- 86. Agribalyse, Agribalyse database. <a href="https://agribalyse.ademe.fr/">https://agribalyse.ademe.fr/</a>.
- 87. Gesundheitswesen, I.f.Q.u.T.i., *Länderbericht Perinatalmedizin: Geburtshilfe. Erfassungsjahr* 2021. 2021.
- 88. Statista. *Bevölkerung Zahl der weiblichen Einwohner in Deutschland nach Altersgruppen am* 31. *Dezember* 2021. 2023 24.03.2023]; Available from: <a href="https://de.statista.com/statistik/daten/studie/1112611/umfrage/weibliche-bevoelkerung-in-deutschland-nach-altersgruppen/">https://de.statista.com/statistik/daten/studie/1112611/umfrage/weibliche-bevoelkerung-in-deutschland-nach-altersgruppen/</a>.
- 89. Kilb, M., et al., Gesundheitliche Auswirkungen einer vegetarischen oder veganen Ernährung bei Kindern der longitudinalen Mutter-Kind-Kohorte PEACHES. 2023.
- 90. Destatis. Familien mit minderjährigen Kindern in der Familie nach Lebensform und Kinderzahl.
  2023 [cited 2023 27.03.2023]; Available from:
  <a href="https://www.destatis.de/DE/Themen/Gesellschaft-Umwelt/Bevoelkerung/Haushalte-Familien/Tabellen/2-5-familien.html">https://www.destatis.de/DE/Themen/Gesellschaft-Umwelt/Bevoelkerung/Haushalte-Familien/Tabellen/2-5-familien.html</a>.
- 91. Destatis, Bevölkerung und Erwerbstätigkeit. Haushalte und Familien. Ergebnisse des Mikrozensus. 2022.
- 92. Mensink, G.B.M., et al., *EsKiMo II Die Ernährungsstudie als KiGGS-Modul*. 2021, Robert Koch-Institut.
- 93. Mensink, G. and M. Burger, *Was isst du? Ein Verzehrshäufigkeitsfragebogen für Kinder und Jugendliche.* Bundesgesundheitsbl Gesundheitsforsch Gesundheitsschutz, 2004. **47**(3).
- 94. Mauz, E., et al., *Neue Daten für Taten. Die Datenerhebung zur KiGGS Welle 2 ist beendet.* Journal of Health Monitoring, 2017. **2**(S3).
- 95. Hoffmann, W., et al., *Guidelines and recommendations for ensuring Good Epidemiological Practice (GEP): a guideline developed by the German Society for Epidemiology.* Eur J Epidemiol, 2019. **34**(3): p. 301-317.
- 96. Schmidt, C.O., et al., *Qualitätsstandards für epidemiologische Kohortenstudien.*Bundesgesundheitsblatt Gesundheitsforschung Gesundheitsschutz, 2018. **61**(1): p. 65-77.

# **Anhang**

# A1 Ablauf der Ernährungserhebung mit der NutriDiary-App



# Anhang A2 Biomarker des Sets 1 (Sofortige Analyse)

| Großes Blutbild | Matrix |
|-----------------------------------------------------------|--------|
| Hämoglobin | Blut |
| Hämatokrit | Blut |
| MCV | Blut |
| MCHC | Blut |
| Erythrozyten | Blut |
| Leukozyten | Blut |
| Lymphozyten | Blut |
| Neutrophile | Blut |
| Basophile | Blut |
| Eosinophile | Blut |
| Thrombozyten | Blut |
| Elektrolyte und Mineralstoffe | |
| Natrium | Blut |
| Kalium | Blut |
| Calcium | Blut |
| Phosphat | Blut |
| Eisen | Blut |
| Magnesium | Blut |
| Leberparameter | |
| Gamma-GT | Blut |
| GOT | Blut |
| GPT | Blut |
| Bilirubin | Blut |
| Blutfette und Entzündungsmarker | |
| Gesamtcholesterin | Blut |
| LDL-Cholesterin | Blut |
| HDL-Cholesterin | Blut |
| Triglyzeride | Blut |
| Hochsensitives C-reaktives Protein | Blut |
| Blutzucker und Diabetesmarker | |
| Nüchternglukose | Blut |
| HbA1c | Blut |
| Nierenparameter | |
| Kreatinin | Blut |
| Harnsäure | Blut |
| 24-Stunden-Urin | |
| Natrium | Urin |
| Kalium | Urin |
| Calcium | Urin |
| Kreatinin | Urin |
| рН | Urin |
| Urin-Teststreifen (Mikroalbumine, Proteinurie, Hämaturie) | Urin |
| Stuhl | |
| pH | Stuhl |

# Anhang A 3 Liste der Biomarker Sets 2 (Spätere Analyse)

Für das Biomarker Set 2 werden die Bioproben für die spätere Analyse gelagert und bei -80°C gelagert. Es sollen Parameter für die Beantwortung verschiedener Fragestellungen analysiert werden:

- Vitamine
- Mineralstoffe
- Spurenelemente
- Schilddrüse
- Herzkreislauf Parameter (Fettsäuren, Homocystein, Apoliloproteine, BNP etc.)
- Knochenstoffwechsel (Osteocalcin, Adinopectin, CTX etc.)
- Entzündung
- Kontaminanten

| Parameter Set 2A | Material | Parameter Set 2A | Material |
|---|---|---|---|
| Lipoprotein(a) | Lithiumheparin | Insulin | Serum |
| NT-proBNP | Lithiumheparin | Osteocalcin | Serum |
| Gesamtprotein | Lithiumheparin | TPO-AK | Serum |
| Harnstoff | Lithiumheparin | Thyreoglobulin | Serum |
| TSH | Lithiumheparin | Thyreoglobulin-AK | Serum |
| fT3 | Lithiumheparin | Ostase | Serum |
| fT4 | Lithiumheparin | Eisen | Lithiumhepa-<br>rin |
| Vitamin B12 | Serum | Ferritin | Lithiumhepa-<br>rin |
| Holo-Transcobalamin | Serum | Transferrin | Lithiumhepa-<br>rin |
| Cystatin C | Serum | Homocystein | EDTA |
| C-Peptid | Serum | Parathormon | EDTA |
| Vitamin D | Serum | | |

| Parameter Set 2B | Material | Parameter Set 2B | Material |
|---|---|---|---|
| Schwermetalle, Me-talloide** | Serum | PINP | Serum |
| PFAS | EDTA-Plasma | Selenoprotein, Selen<br>Mangan, Kupfer, Ceruloplasmin | Serum |
| Dioxin, PCBs | EDTA-Plasma | Vitamine: A, B1, B2, B3, B5, B6, D, E, H, K, Folat | EDTA-<br>Plasma |
| Mykotoxine | Serum | Untargeted Metabolomics | EDTA-<br>Plasma |
| Inflammatorische Marker (z.B. Adiponektin, Omentin) | EDTA-Plasma | Targeted Metabolomics | Serum/E-<br>Plasma |
| Inflammatorische Marker | Serum | Süßungsmittel | 24 h S Urin |
| Ak Hep E | Serum | Weichmacher | 24 h S Urin |
| Ak Toxoplasmose | Serum | Mercaptursäuren*** | 24 h S Urin |

| Ak Kryptosporidien | Serum | Albumin, Natrium, Magnesium,<br>Phosphat, Kalium, Eisen, Os-<br>molarität, Jod | 24 h S Urin |
|---|---|---|---|
| BMMF Bovine Meat +Milk Factors | Serum | Knochenmetabolismusmarker | 24 h S Urin |
| FGF23 /Alpha Klotho | EDTA-Plasma | Untargeted Metabolomics | 24 h S Urin |
| ApoA1, Apo B | Serum | Hämoglobinaddukte | Ery-Aufar-<br>beitung |
| Oxidativer Stress<br>(z.B. Malondialdehyd-modifiz.<br>LDL) | Serum | Fettsäuren | Ery-Aufar-<br>beitung |
| RANKL/Osteoprotegerin | Serum | Methylierung | EDTA-Voll-<br>blut |
| B-cross-Laps (CTX) /Desox-<br>ypyridinolin-Crosslinks<br>(DPD) PINP | Serum | Aminosäuren* | EDTA-<br>Plasma |

<sup>\*</sup> Aminosäuren: Histidin, Isoleucin, Leucin, Lysin, Methionin, Phenylalanin, Threonin, Tryptophan, Valin, Alanin, Arginin, Asparagin, Asparaginsäure, Cystein, Glutamin, Glycin, Prolin, Serin, Tyrosin
\*\* Kontaminanten: Metalle / Metalloide (z.B. Cadmium, Arsenspezies), PFAS, Dioxin/PCBs (gepoolte Proben), Mykotoxine, hitzebedingte Kontaminanten (Hämoglobinaddukte), Fettsäuren
\*\*\* Spezifische Merkaptursäuren von hitzebedingten Kontaminanten, MCPD